CLINICAL TRIAL: NCT01559259
Title: EVALUATION OF THE EFFICACY OF NOVEL IBUPROFEN ACETAMINOPHEN COMBINATION FORMULATIONS IN THE TREATMENT OF POST-SURGICAL DENTAL PAIN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B5061001
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Results first posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Pain
Keywords: ibuprofen; acetaminophen; pain; molar extraction
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ibuprofen/acetaminophen (lower dose) (Experimental)
  Interventions: Drug: Ibuprofen/acetaminophen
- Ibuprofen/acetaminophen (middle dose) (Experimental)
  Interventions: Drug: Ibuprofen/acetaminophen
- Ibuprofen/acetaminophen (high dose) (Experimental)
  Interventions: Drug: Ibuprofen/acetaminophen
- Ibuprofen (Active Comparator)
  Interventions: Drug: Ibuprofen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen/acetaminophen — Two caplets of ibuprofen 100 mg plus acetaminophen 250 mg
  Arms: Ibuprofen/acetaminophen (lower dose)
Drug: Ibuprofen/acetaminophen — Two caplets of ibuprofen 125 mg plus acetaminophen 250 mg
  Arms: Ibuprofen/acetaminophen (middle dose)
Drug: Ibuprofen/acetaminophen — Two caplets of ibuprofen 150 mg plus acetaminophen 250 mg
  Arms: Ibuprofen/acetaminophen (high dose)
Drug: Ibuprofen — Two caplets of ibuprofen 200 mg
  Arms: Ibuprofen
Drug: Placebo — Two caplets of placebo
  Arms: Placebo

SUMMARY:
This study will determine the overall analgesic efficacy of three different fixed dose ibuprofen plus acetaminophen formulations compared to ibuprofen alone and to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 16 to 40 years of age
* Moderate to severe post-operative pain following surgical extraction of three or more third molar teeth

Exclusion Criteria:

* Presence of history of significant hepatic, renal, endocrine, cardiovascular, neurological, psychiatric, gastrointestinal, pulmonary, hematologic or metabolic disorder
* Pregnant or breastfeeding females

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 394 (Actual)
Dates: Start 2012-04-10 (Actual); Primary Completion 2012-09-13 (Actual); Study Completion 2012-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Jean Brown Research, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kellstein D, Leyva R. Evaluation of Fixed-Dose Combinations of Ibuprofen and Acetaminophen in the Treatment of Postsurgical Dental Pain: A Pilot, Dose-Ranging, Randomized Study. Drugs R D. 2020 Sep;20(3):237-247. doi: 10.1007/s40268-020-00310-7. PMID 32506309
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5061001&StudyName=Evaluation%20of%20the%20Efficacy%20of%20Novel%20Ibuprofen%20Acetaminophen%20Combination%20Formulations%20in%20the%20Treatment%20of%20Post-surgical%20Dental%20Pain

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received Placebo as single oral dose caplets during the 12 hours study.
- Ibuprofen 200 mg + Acetaminophen 500 mg: Participants received a single oral dose of a fixed dose combination of ibuprofen 200 milligram (mg) and acetaminophen 500 mg caplets during the 12 hours study.
- Ibuprofen 250 mg + Acetaminophen 500 mg: Participants received a single oral dose of a fixed dose combination of ibuprofen 250 mg and acetaminophen 500 mg caplets during the 12 hours study.
- Ibuprofen 300 mg + Acetaminophen 500 mg: Participants received a single oral dose of a fixed dose combination of ibuprofen 300 mg and acetaminophen 500 mg caplets during the 12 hours study.
- Ibuprofen 400 mg: Participants received single oral dose of ibuprofen 400 mg caplets during the 12 hours study.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Started | 30 | 90 | 93 | 89 | 92
Completed | 30 | 89 | 92 | 88 | 92
Not Completed | 0 | 1 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication and provided a baseline assessment.
Groups:
- Ibuprofen 200 mg + Acetaminophen 500 mg: Participants received a single oral dose of a fixed dose combination of ibuprofen 200 mg and acetaminophen 500 mg caplets during the 12 hours study.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg | Total
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (2.6) | 17.7 (1.8) | 18.4 (2.1) | 17.8 (1.8) | 18.4 (1.9) | 18.1 (2.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 46 | 50 | 43 | 46 | 200
  Male | 15 | 44 | 43 | 46 | 46 | 194

OUTCOME MEASURES:

1. Primary Outcome: Time-Weighted Sum of Pain Relief Rating and Pain Intensity Difference Scores From 0 to 8 Hours (SPRID 0-8)
Description: SPRID4:Time-weighted sum of pain relief rating (PRR) and pain intensity difference (PID) based on 4 point categorical severity rating scale (PRID) over 8 hours.SPRID 0-8 score range:-8 (worst score) to 56 (best score).PRID: sum of PRR and PID at each time point.PRID score range:-1= worst score to 7= best score.PID4 was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [none] to 3 [severe]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 = severe pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -1 (worst score) to 3 (best score).PRR assessed on 5-point categorical scale with range:0 =no relief to 4 =complete relief.
Time Frame: From 0 hour up to 8 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale | 5.0 (13.2) | 30.8 (12.7) | 29.6 (15.6) | 31.7 (14.6) | 28.8 (15.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; Treatment difference and 95 percent (%) Confidence interval (CI) were based on Least square mean (LSM) from analysis of variance (ANOVA) with treatment, baseline categorical pain severity rating (PSR), gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; Least Square (LS) Mean difference = 26.28, 95% CI 2-sided [20.33 to 32.22]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 24.37, 95% CI 2-sided [18.44 to 30.29]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 27.48, 95% CI 2-sided [21.53 to 33.42]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 24.85, 95% CI 2-sided [18.93 to 30.78]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.501, ANOVA; LS Mean difference = 1.42, 95% CI 2-sided [-2.73 to 5.58]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.817, ANOVA; LS Mean difference = -0.49, 95% CI 2-sided [-4.61 to 3.64]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.216, ANOVA; LS Mean difference = 2.62, 95% CI 2-sided [-1.53 to 6.78]

2. Secondary Outcome: Time to Onset of Meaningful Pain Relief
Description: Participants evaluated time to meaningful relief by stopping a second stopwatch labelled as "meaningful relief" at the moment they first began to experience meaningful relief. Stopwatch was active up to 12 hours after dosing or until stopped by participant, or participant became treatment failure prior to depressing the second stopwatch. Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: From 0 hour up to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
minutes | NA [NA to NA] — Median was not analysed as median time to meaningful relief was greater than (>) 720 minutes/12 hours) for placebo group and therefore 95% CI was not estimable. | 44.5 [37.0 to 55.0] | 54.1 [44.7 to 73.6] | 45.9 [42.2 to 57.2] | 56.2 [52.0 to 77.0]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; Hazard ratio (HR) and corresponding 95% CI were calculated based on the Wald statistic from the proportional hazards (PH) model with treatment, baseline categorical PSR and gender terms used as covariates; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 12.69, 95% CI 2-sided [5.52 to 29.19]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 10.02, 95% CI 2-sided [4.36 to 23.02]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 11.66, 95% CI 2-sided [5.07 to 26.83]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 8.60, 95% CI 2-sided [3.74 to 19.77]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.014, Proportional hazards model; Hazard Ratio (HR) = 1.48, 95% CI 2-sided [1.08 to 2.02]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.332, Proportional hazards model; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.86 to 1.59]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.056, Proportional hazards model; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [0.99 to 1.85]

3. Secondary Outcome: Time to Confirmed First Perceptible Relief
Description: Participants evaluated the time to first perceptible relief (confirmed by meaningful relief) by stopping the first stopwatch labelled 'first perceptible relief' at the moment they first began to experience any pain relief, if the participant also achieved meaningful relief by the end of the study. Stopwatch was active up to 12 hours after dosing or until stopped by the participant, or until the participant dropped out due to treatment failure (defined as participant taking rescue medication, or discontinuing due to lack of efficacy) prior to depressing the first stopwatch or until the time of withdrawal (discontinuation).
Time Frame: From 0 hour up to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
minutes | NA [NA to NA] — Median was not analysed as median time to confirmed first perceptible relief was >720 minutes (>12 hours) for placebo group and therefore 95% CI was not estimable. | 18.5 [15.7 to 23.0] | 22.8 [19.9 to 27.4] | 18.5 [15.7 to 21.8] | 24.9 [21.6 to 28.7]
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical PSR and gender terms used as covariates; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 12.10, 95% CI 2-sided [5.24 to 27.91]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 8.88, 95% CI 2-sided [3.86 to 20.44]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 11.47, 95% CI 2-sided [4.98 to 26.42]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Proportional hazards model; Hazard Ratio (HR) = 8.11, 95% CI 2-sided [3.52 to 18.68]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.012, Proportional hazards model; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.09 to 2.04]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.570, Proportional hazards model; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.80 to 1.49]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.030, Proportional hazards model; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [1.03 to 1.93]

4. Secondary Outcome: Pain Relief Rating Score (PRR)
Description: Participants answered a question: "how much relief do you have from your starting pain? on a 5-point categorical pain relief rating scale. Scale ranges from 0= no relief to 4= complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0.25 hour | 0.2 (0.4) | 0.6 (0.8) | 0.5 (0.8) | 0.7 (0.9) | 0.4 (0.6)
  0.5 hour | 0.3 (0.5) | 1.7 (1.0) | 1.5 (1.2) | 1.6 (1.1) | 1.1 (0.9)
  1 hour | 0.4 (0.6) | 2.5 (1.1) | 2.3 (1.1) | 2.5 (1.2) | 2.1 (1.1)
  1.5 hour | 0.4 (0.8) | 2.8 (0.9) | 2.6 (1.1) | 2.8 (1.0) | 2.5 (1.2)
  2 hour | 0.4 (0.8) | 2.9 (1.0) | 2.7 (1.2) | 2.9 (1.1) | 2.6 (1.3)
  3 hour | 0.5 (1.0) | 2.9 (1.0) | 2.8 (1.2) | 3.0 (1.2) | 2.7 (1.3)
  4 hour | 0.5 (1.1) | 2.9 (1.0) | 2.7 (1.3) | 2.9 (1.2) | 2.7 (1.4)
  5 hour | 0.5 (1.1) | 2.7 (1.1) | 2.6 (1.3) | 2.8 (1.3) | 2.6 (1.4)
  6 hour | 0.6 (1.2) | 2.5 (1.3) | 2.4 (1.4) | 2.7 (1.4) | 2.4 (1.5)
  7 hour | 0.6 (1.2) | 2.1 (1.4) | 2.2 (1.4) | 2.3 (1.4) | 2.1 (1.5)
  8 hour | 0.6 (1.2) | 1.7 (1.5) | 1.9 (1.4) | 1.9 (1.5) | 1.9 (1.5)
  9 hour | 0.6 (1.2) | 1.4 (1.5) | 1.5 (1.4) | 1.7 (1.5) | 1.7 (1.5)
  10 hour | 0.6 (1.2) | 1.2 (1.4) | 1.2 (1.3) | 1.5 (1.5) | 1.4 (1.5)
  11 hour | 0.6 (1.3) | 0.9 (1.4) | 1.0 (1.3) | 1.3 (1.4) | 1.3 (1.5)
  12 hour | 0.6 (1.3) | 0.8 (1.3) | 0.9 (1.2) | 1.1 (1.3) | 1.2 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.25 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean difference = 0.39, 95% CI 2-sided [0.08 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.038, ANOVA; LS Mean difference = 0.33, 95% CI 2-sided [0.02 to 0.64]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean difference = 0.48, 95% CI 2-sided [0.17 to 0.79]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.155, ANOVA; LS Mean difference = 0.23, 95% CI 2-sided [-0.09 to 0.54]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.135, ANOVA; LS Mean difference = 0.17, 95% CI 2-sided [-0.05 to 0.39]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.350, ANOVA; LS Mean difference = 0.10, 95% CI 2-sided [-0.11 to 0.32]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean difference = 0.25, 95% CI 2-sided [0.03 to 0.47]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.5 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.33, 95% CI 2-sided [0.90 to 1.77]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.26, 95% CI 2-sided [0.83 to 1.70]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean difference = 1.35, 95% CI 2-sided [0.91 to 1.78]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.87, 95% CI 2-sided [0.43 to 1.30]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean difference = 0.47, 95% CI 2-sided [0.16 to 0.77]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.010, ANOVA; LS Mean difference = 0.40, 95% CI 2-sided [0.10 to 0.70]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 0.48, 95% CI 2-sided [0.18 to 0.79]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 1 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.12, 95% CI 2-sided [1.66 to 2.58]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.96, 95% CI 2-sided [1.50 to 2.42]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.14, 95% CI 2-sided [1.67 to 2.60]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.74, 95% CI 2-sided [1.28 to 2.20]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.022, ANOVA; LS Mean difference = 0.38, 95% CI 2-sided [0.05 to 0.70]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.181, ANOVA; LS Mean difference = 0.22, 95% CI 2-sided [-0.10 to 0.54]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.016, ANOVA; LS Mean difference = 0.40, 95% CI 2-sided [0.07 to 0.72]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 1.5 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.43, 95% CI 2-sided [1.98 to 2.88]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.17, 95% CI 2-sided [1.72 to 2.62]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.46, 95% CI 2-sided [2.01 to 2.91]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.13, 95% CI 2-sided [1.68 to 2.58]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.065, ANOVA; LS Mean difference = 0.30, 95% CI 2-sided [-0.02 to 0.61]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.817, ANOVA; LS Mean difference = 0.04, 95% CI 2-sided [-0.28 to 0.35]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.043, ANOVA; LS Mean difference = 0.33, 95% CI 2-sided [0.01 to 0.64]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 2 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.53, 95% CI 2-sided [2.06 to 3.01]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.34, 95% CI 2-sided [1.87 to 2.82]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.63, 95% CI 2-sided [2.15 to 3.11]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.36, 95% CI 2-sided [1.89 to 2.84]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.312, ANOVA; LS Mean difference = 0.17, 95% CI 2-sided [-0.16 to 0.51]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.910, ANOVA; LS Mean difference = -0.02, 95% CI 2-sided [-0.35 to 0.31]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.113, ANOVA; LS Mean difference = 0.27, 95% CI 2-sided [-0.06 to 0.60]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 3 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.48, 95% CI 2-sided [1.98 to 2.97]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.25, 95% CI 2-sided [1.76 to 2.75]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.51, 95% CI 2-sided [2.02 to 3.01]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.35, 95% CI 2-sided [1.86 to 2.85]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.482, ANOVA; LS Mean difference = 0.12, 95% CI 2-sided [-0.22 to 0.47]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.573, ANOVA; LS Mean difference = -0.10, 95% CI 2-sided [-0.44 to 0.24]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.368, ANOVA; LS Mean difference = 0.16, 95% CI 2-sided [-0.19 to 0.50]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 4 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.40, 95% CI 2-sided [1.88 to 2.91]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.17, 95% CI 2-sided [1.66 to 2.68]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.44, 95% CI 2-sided [1.93 to 2.96]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.23, 95% CI 2-sided [1.72 to 2.74]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.352, ANOVA; LS Mean difference = 0.17, 95% CI 2-sided [-0.19 to 0.53]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.771, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.41 to 0.30]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.235, ANOVA; LS Mean difference = 0.22, 95% CI 2-sided [-0.14 to 0.58]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 5 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.32, 95% CI 2-sided [1.79 to 2.86]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.05, 95% CI 2-sided [1.52 to 2.58]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.37, 95% CI 2-sided [1.83 to 2.90]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.20, 95% CI 2-sided [1.66 to 2.73]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.510, ANOVA; LS Mean difference = 0.13, 95% CI 2-sided [-0.25 to 0.50]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.442, ANOVA; LS Mean difference = -0.15, 95% CI 2-sided [-0.52 to 0.23]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.372, ANOVA; LS Mean difference = 0.17, 95% CI 2-sided [-0.20 to 0.54]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 6 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.97, 95% CI 2-sided [1.39 to 2.55]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.82, 95% CI 2-sided [1.25 to 2.40]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.15, 95% CI 2-sided [1.57 to 2.72]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.87, 95% CI 2-sided [1.30 to 2.45]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.639, ANOVA; LS Mean difference = 0.10, 95% CI 2-sided [-0.31 to 0.50]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.803, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.45 to 0.35]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.184, ANOVA; LS Mean difference = 0.27, 95% CI 2-sided [-0.13 to 0.67]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 7 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.67, 95% CI 2-sided [1.07 to 2.26]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.58, 95% CI 2-sided [0.99 to 2.17]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.84, 95% CI 2-sided [1.25 to 2.43]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.69, 95% CI 2-sided [1.10 to 2.28]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.910, ANOVA; LS Mean difference = -0.02, 95% CI 2-sided [-0.44 to 0.39]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.607, ANOVA; LS Mean difference = -0.11, 95% CI 2-sided [-0.52 to 0.30]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.484, ANOVA; LS Mean difference = 0.15, 95% CI 2-sided [-0.27 to 0.56]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 8 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.25, 95% CI 2-sided [0.64 to 1.86]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.36, 95% CI 2-sided [0.75 to 1.97]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.38, 95% CI 2-sided [0.77 to 1.99]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.50, 95% CI 2-sided [0.89 to 2.10]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.256, ANOVA; LS Mean difference = -0.25, 95% CI 2-sided [-0.67 to 0.18]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.526, ANOVA; LS Mean difference = -0.14, 95% CI 2-sided [-0.56 to 0.29]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.602, ANOVA; LS Mean difference = -0.11, 95% CI 2-sided [-0.54 to 0.31]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 9 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 0.95, 95% CI 2-sided [0.34 to 1.56]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean difference = 0.98, 95% CI 2-sided [0.38 to 1.59]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.25, 95% CI 2-sided [0.65 to 1.86]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.22, 95% CI 2-sided [0.61 to 1.82]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.224, ANOVA; LS Mean difference = -0.26, 95% CI 2-sided [-0.69 to 0.16]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.283, ANOVA; LS Mean difference = -0.23, 95% CI 2-sided [-0.65 to 0.19]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.860, ANOVA; LS Mean difference = 0.04, 95% CI 2-sided [-0.39 to 0.46]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 10 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.038, ANOVA; LS Mean difference = 0.63, 95% CI 2-sided [0.03 to 1.22]
Statistical Analysis 86: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean difference = 0.65, 95% CI 2-sided [0.06 to 1.24]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.03, 95% CI 2-sided [0.43 to 1.62]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 0.95, 95% CI 2-sided [0.36 to 1.54]
Statistical Analysis 89: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.129, ANOVA; LS Mean difference = -0.32, 95% CI 2-sided [-0.74 to 0.09]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.154, ANOVA; LS Mean difference = -0.30, 95% CI 2-sided [-0.71 to 0.11]
Statistical Analysis 91: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.714, ANOVA; LS Mean difference = 0.08, 95% CI 2-sided [-0.34 to 0.49]
Statistical Analysis 92: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 11 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.217, ANOVA; LS Mean difference = 0.37, 95% CI 2-sided [-0.22 to 0.96]
Statistical Analysis 93: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.136, ANOVA; LS Mean difference = 0.45, 95% CI 2-sided [-0.14 to 1.03]
Statistical Analysis 94: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.010, ANOVA; LS Mean difference = 0.78, 95% CI 2-sided [0.19 to 1.37]
Statistical Analysis 95: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.006, ANOVA; LS Mean difference = 0.83, 95% CI 2-sided [0.24 to 1.41]
Statistical Analysis 96: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean difference = -0.45, 95% CI 2-sided [-0.87 to -0.04]
Statistical Analysis 97: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.070, ANOVA; LS Mean difference = -0.38, 95% CI 2-sided [-0.79 to 0.03]
Statistical Analysis 98: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.822, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.46 to 0.37]
Statistical Analysis 99: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 12 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.327, ANOVA; LS Mean difference = 0.28, 95% CI 2-sided [-0.28 to 0.83]
Statistical Analysis 100: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.224, ANOVA; LS Mean difference = 0.34, 95% CI 2-sided [-0.21 to 0.89]
Statistical Analysis 101: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.025, ANOVA; LS Mean difference = 0.63, 95% CI 2-sided [0.08 to 1.19]
Statistical Analysis 102: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.012, ANOVA; LS Mean difference = 0.70, 95% CI 2-sided [0.15 to 1.25]
Statistical Analysis 103: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.030, ANOVA; LS Mean difference = -0.43, 95% CI 2-sided [-0.81 to -0.04]
Statistical Analysis 104: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.064, ANOVA; LS Mean difference = -0.36, 95% CI 2-sided [-0.75 to 0.02]
Statistical Analysis 105: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.721, ANOVA; LS Mean difference = -0.07, 95% CI 2-sided [-0.46 to 0.32]

5. Secondary Outcome: Pain Intensity Difference on 4-Point Categorical Scale (PID4)
Description: PID4: baseline pain severity score minus pain severity score at a given time point. Pain intensity was assessed on a 4-point categorical pain severity rating scale. PID4 was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [no pain] to 3 [worst possible pain]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID4: -1 (worst score) to 3 (best score).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0.25 hour | 0.1 (0.3) | 0.3 (0.6) | 0.2 (0.4) | 0.3 (0.6) | 0.2 (0.4)
  0.5 hour | 0.1 (0.4) | 0.9 (0.8) | 0.7 (0.8) | 0.8 (0.8) | 0.5 (0.7)
  1 hour | 0.1 (0.6) | 1.5 (0.9) | 1.2 (0.8) | 1.4 (0.9) | 1.1 (0.9)
  1.5 hour | 0.1 (0.7) | 1.6 (0.8) | 1.5 (1.0) | 1.6 (0.9) | 1.4 (0.9)
  2 hour | 0.0 (0.7) | 1.7 (0.9) | 1.6 (1.0) | 1.7 (0.9) | 1.5 (0.9)
  3 hour | 0.1 (0.8) | 1.7 (0.9) | 1.6 (1.0) | 1.7 (1.0) | 1.6 (1.0)
  4 hour | 0.1 (0.9) | 1.7 (0.9) | 1.6 (1.1) | 1.7 (0.9) | 1.6 (1.0)
  5 hour | 0.1 (0.9) | 1.6 (0.9) | 1.5 (1.1) | 1.6 (1.0) | 1.5 (1.0)
  6 hour | 0.2 (0.9) | 1.4 (1.0) | 1.4 (1.1) | 1.6 (1.1) | 1.3 (1.0)
  7 hour | 0.2 (0.9) | 1.2 (1.0) | 1.2 (1.1) | 1.3 (1.1) | 1.2 (1.0)
  8 hour | 0.2 (0.9) | 0.9 (1.0) | 1.0 (1.0) | 1.0 (1.0) | 1.0 (1.1)
  9 hour | 0.2 (0.9) | 0.8 (1.0) | 0.7 (1.0) | 0.8 (0.9) | 0.8 (1.0)
  10 hour | 0.2 (1.0) | 0.6 (0.9) | 0.6 (0.9) | 0.7 (0.9) | 0.7 (1.0)
  11 hour | 0.2 (1.0) | 0.5 (1.0) | 0.5 (0.9) | 0.6 (0.9) | 0.6 (0.9)
  12 hour | 0.3 (1.1) | 0.3 (0.8) | 0.4 (0.8) | 0.4 (0.8) | 0.5 (0.8)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.033, ANOVA; LS mean difference = 0.22, 95% CI 2-sided [0.02 to 0.42]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.224, ANOVA; LS Mean difference = 0.13, 95% CI 2-sided [-0.08 to 0.33]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean difference = 0.23, 95% CI 2-sided [0.03 to 0.44]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.501, ANOVA; LS Mean difference = 0.07, 95% CI 2-sided [-0.13 to 0.27]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.036, ANOVA; LS Mean difference = 0.15, 95% CI 2-sided [0.01 to 0.29]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.435, ANOVA; LS Mean difference = 0.06, 95% CI 2-sided [-0.08 to 0.20]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.023, ANOVA; LS Mean difference = 0.16, 95% CI 2-sided [0.02 to 0.31]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.82, 95% CI 2-sided [0.52 to 1.12]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.67, 95% CI 2-sided [0.37 to 0.97]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.74, 95% CI 2-sided [0.45 to 1.04]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean difference = 0.45, 95% CI 2-sided [0.16 to 0.75]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.37, 95% CI 2-sided [0.16 to 0.58]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.039, ANOVA; LS Mean difference = 0.22, 95% CI 2-sided [0.01 to 0.42]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.006, ANOVA; LS Mean difference = 0.29, 95% CI 2-sided [0.08 to 0.50]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.33, 95% CI 2-sided [1.01 to 1.65]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.17, 95% CI 2-sided [0.85 to 1.49]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.35, 95% CI 2-sided [1.03 to 1.67]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.04, 95% CI 2-sided [0.72 to 1.36]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.011, ANOVA; LS Mean difference = 0.29, 95% CI 2-sided [0.07 to 0.52]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.267, ANOVA; LS Mean difference = 0.13, 95% CI 2-sided [-0.10 to 0.35]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.007, ANOVA; LS Mean difference = 0.31, 95% CI 2-sided [0.09 to 0.53]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.57, 95% CI 2-sided [1.24 to 1.89]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.38, 95% CI 2-sided [1.06 to 1.70]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.57, 95% CI 2-sided [1.25 to 1.90]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.35, 95% CI 2-sided [1.02 to 1.67]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.056, ANOVA; LS Mean difference = 0.22, 95% CI 2-sided [-0.01 to 0.45]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.759, ANOVA; LS Mean difference = 0.04, 95% CI 2-sided [-0.19 to 0.26]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.051, ANOVA; LS Mean difference = 0.23, 95% CI 2-sided [-0.00 to 0.45]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.64, 95% CI 2-sided [1.30 to 1.98]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.52, 95% CI 2-sided [1.18 to 1.85]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.71, 95% CI 2-sided [1.37 to 2.05]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.52, 95% CI 2-sided [1.19 to 1.86]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.342, ANOVA; LS Mean difference = 0.11, 95% CI 2-sided [-0.12 to 0.35]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.943, ANOVA; LS Mean difference = -0.01, 95% CI 2-sided [-0.24 to 0.23]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.126, ANOVA; LS Mean difference = 0.18, 95% CI 2-sided [-0.05 to 0.42]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.63, 95% CI 2-sided [1.27 to 1.98]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.50, 95% CI 2-sided [1.15 to 1.86]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.64, 95% CI 2-sided [1.29 to 2.00]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.53, 95% CI 2-sided [1.18 to 1.89]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.453, ANOVA; LS Mean difference = 0.10, 95% CI 2-sided [-0.15 to 0.34]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.816, ANOVA; LS Mean difference = -0.03, 95% CI 2-sided [-0.28 to 0.22]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.384, ANOVA; LS Mean difference = 0.11, 95% CI 2-sided [-0.14 to 0.36]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.55, 95% CI 2-sided [1.19 to 1.91]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.46, 95% CI 2-sided [1.10 to 1.82]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.61, 95% CI 2-sided [1.25 to 1.97]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.46, 95% CI 2-sided [1.10 to 1.82]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.483, ANOVA; LS Mean difference = 0.09, 95% CI 2-sided [-0.16 to 0.34]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.991, ANOVA; LS Mean difference = 0.00, 95% CI 2-sided [-0.25 to 0.25]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.228, ANOVA; LS Mean difference = 0.16, 95% CI 2-sided [-0.10 to 0.41]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.48, 95% CI 2-sided [1.10 to 1.85]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.32, 95% CI 2-sided [0.94 to 1.69]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.53, 95% CI 2-sided [1.15 to 1.90]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.40, 95% CI 2-sided [1.03 to 1.78]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.587, ANOVA; LS Mean difference = 0.07, 95% CI 2-sided [-0.19 to 0.33]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.517, ANOVA; LS Mean difference = -0.09, 95% CI 2-sided [-0.35 to 0.17]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.360, ANOVA; LS Mean difference = 0.12, 95% CI 2-sided [-0.14 to 0.38]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.20, 95% CI 2-sided [0.81 to 1.60]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.17, 95% CI 2-sided [0.78 to 1.57]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.36, 95% CI 2-sided [0.97 to 1.76]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.17, 95% CI 2-sided [0.77 to 1.56]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.811, ANOVA; LS Mean difference = 0.03, 95% CI 2-sided [-0.24 to 0.31]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.977, ANOVA; LS Mean difference = 0.00, 95% CI 2-sided [-0.27 to 0.28]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.164, ANOVA; LS Mean difference = 0.20, 95% CI 2-sided [-0.08 to 0.47]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.03, 95% CI 2-sided [0.63 to 1.43]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.00, 95% CI 2-sided [0.60 to 1.40]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.15, 95% CI 2-sided [0.75 to 1.56]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.06, 95% CI 2-sided [0.66 to 1.46]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.846, ANOVA; LS Mean difference = -0.03, 95% CI 2-sided [-0.31 to 0.25]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.702, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.33 to 0.23]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.496, ANOVA; LS Mean difference = 0.10, 95% CI 2-sided [-0.18 to 0.38]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.81, 95% CI 2-sided [0.41 to 1.22]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.81, 95% CI 2-sided [0.40 to 1.21]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.86, 95% CI 2-sided [0.46 to 1.26]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.92, 95% CI 2-sided [0.52 to 1.33]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.441, ANOVA; LS Mean difference = -0.11, 95% CI 2-sided [-0.39 to 0.17]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.408, ANOVA; LS Mean difference = -0.12, 95% CI 2-sided [-0.40 to 0.16]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.652, ANOVA; LS Mean difference = -0.06, 95% CI 2-sided [-0.35 to 0.22]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean difference = 0.61, 95% CI 2-sided [0.21 to 1.02]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.007, ANOVA; LS Mean difference = 0.55, 95% CI 2-sided [0.15 to 0.95]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.69, 95% CI 2-sided [0.29 to 1.10]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.70, 95% CI 2-sided [0.29 to 1.10]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.567, ANOVA; LS Mean difference = -0.08, 95% CI 2-sided [-0.36 to 0.20]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.315, ANOVA; LS Mean difference = -0.14, 95% CI 2-sided [-0.42 to 0.14]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.997, ANOVA; LS Mean difference = 0.00, 95% CI 2-sided [-0.28 to 0.28]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.056, ANOVA; LS Mean difference = 0.38, 95% CI 2-sided [-0.01 to 0.77]
Statistical Analysis 86: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.047, ANOVA; LS Mean difference = 0.39, 95% CI 2-sided [0.01 to 0.78]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.005, ANOVA; LS Mean difference = 0.56, 95% CI 2-sided [0.17 to 0.95]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.007, ANOVA; LS Mean difference = 0.53, 95% CI 2-sided [0.14 to 0.92]
Statistical Analysis 89: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.276, ANOVA; LS Mean difference = -0.15, 95% CI 2-sided [-0.42 to 0.12]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.318, ANOVA; LS Mean difference = -0.14, 95% CI 2-sided [-0.41 to 0.13]
Statistical Analysis 91: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.849, ANOVA; LS Mean difference = 0.03, 95% CI 2-sided [-0.25 to 0.30]
Statistical Analysis 92: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.138, ANOVA; LS Mean difference = 0.29, 95% CI 2-sided [-0.09 to 0.66]
Statistical Analysis 93: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.111, ANOVA; LS Mean difference = 0.31, 95% CI 2-sided [-0.07 to 0.68]
Statistical Analysis 94: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean difference = 0.42, 95% CI 2-sided [0.04 to 0.79]
Statistical Analysis 95: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.011, ANOVA; LS Mean difference = 0.49, 95% CI 2-sided [0.11 to 0.87]
Statistical Analysis 96: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.135, ANOVA; LS Mean difference = -0.20, 95% CI 2-sided [-0.47 to 0.06]
Statistical Analysis 97: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.175, ANOVA; LS Mean difference = -0.18, 95% CI 2-sided [-0.44 to 0.08]
Statistical Analysis 98: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.590, ANOVA; LS Mean difference = -0.07, 95% CI 2-sided [-0.34 to 0.19]
Statistical Analysis 99: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.402, ANOVA; LS Mean difference = 0.15, 95% CI 2-sided [-0.20 to 0.49]
Statistical Analysis 100: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.261, ANOVA; LS Mean difference = 0.20, 95% CI 2-sided [-0.15 to 0.54]
Statistical Analysis 101: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.134, ANOVA; LS Mean difference = 0.26, 95% CI 2-sided [-0.08 to 0.61]
Statistical Analysis 102: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean difference = 0.38, 95% CI 2-sided [0.03 to 0.72]
Statistical Analysis 103: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.061, ANOVA; LS Mean difference = -0.23, 95% CI 2-sided [-0.47 to 0.01]
Statistical Analysis 104: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.138, ANOVA; LS Mean difference = -0.18, 95% CI 2-sided [-0.42 to 0.06]
Statistical Analysis 105: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.353, ANOVA; LS Mean difference = -0.11, 95% CI 2-sided [-0.35 to 0.13]

6. Secondary Outcome: Pain Intensity Difference on 11-Point Numerical Scale (PID11)
Description: PID11: baseline pain severity score minus pain severity score at a given time point. Pain intensity was assessed on an 11-point numerical pain severity rating scale. PID11 was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID11: -5 (worst score) to 10 (best score).
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0.25 hour | 0.1 (0.6) | 1.0 (1.6) | 0.8 (1.3) | 0.9 (1.6) | 0.4 (1.0)
  0.5 hour | 0.2 (1.1) | 3.0 (2.3) | 2.5 (2.3) | 2.6 (2.3) | 1.7 (1.8)
  1 hour | 0.1 (1.4) | 4.7 (2.5) | 4.2 (2.6) | 4.5 (2.4) | 3.8 (2.6)
  1.5 hour | 0.0 (1.7) | 5.3 (2.4) | 5.0 (2.8) | 5.3 (2.4) | 4.6 (2.7)
  2 hour | -0.1 (1.8) | 5.5 (2.5) | 5.3 (3.0) | 5.6 (2.5) | 5.0 (2.8)
  3 hour | 0.1 (2.2) | 5.7 (2.5) | 5.5 (3.0) | 5.7 (2.7) | 5.2 (2.9)
  4 hour | 0.3 (2.5) | 5.5 (2.5) | 5.4 (3.1) | 5.6 (2.7) | 5.1 (3.0)
  5 hour | 0.2 (2.4) | 5.3 (2.6) | 5.1 (3.2) | 5.3 (3.0) | 4.9 (3.0)
  6 hour | 0.4 (2.6) | 4.6 (2.9) | 4.8 (3.3) | 5.0 (3.1) | 4.4 (3.2)
  7 hour | 0.3 (2.5) | 3.9 (2.9) | 4.2 (3.2) | 4.2 (3.1) | 3.9 (3.2)
  8 hour | 0.3 (2.6) | 3.1 (3.0) | 3.5 (3.2) | 3.2 (3.0) | 3.5 (3.2)
  9 hour | 0.5 (2.8) | 2.5 (3.0) | 2.7 (3.1) | 2.8 (3.0) | 2.9 (3.0)
  10 hour | 0.6 (3.0) | 1.9 (2.8) | 2.1 (3.0) | 2.5 (2.9) | 2.5 (3.0)
  11 hour | 0.6 (2.9) | 1.6 (2.8) | 1.7 (2.9) | 2.0 (2.6) | 2.2 (2.9)
  12 hour | 0.7 (3.2) | 1.1 (2.4) | 1.5 (2.6) | 1.7 (2.5) | 1.9 (2.6)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.25 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.006, ANOVA; LS mean difference = 0.88, 95% CI 2-sided [0.25 to 1.51]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.030, ANOVA; LS Mean difference = 0.69, 95% CI 2-sided [0.07 to 1.31]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.012, ANOVA; LS Mean difference = 0.81, 95% CI 2-sided [0.17 to 1.44]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.237, ANOVA; LS Mean difference = 0.38, 95% CI 2-sided [-0.25 to 1.01]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.024, ANOVA; LS Mean difference = 0.50, 95% CI 2-sided [0.07 to 0.93]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.150, ANOVA; LS Mean difference = 0.31, 95% CI 2-sided [-0.11 to 0.73]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.054, ANOVA; LS Mean difference = 0.43, 95% CI 2-sided [-0.01 to 0.86]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.5 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.89, 95% CI 2-sided [1.92 to 3.85]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.52, 95% CI 2-sided [1.56 to 3.47]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.51, 95% CI 2-sided [1.54 to 3.47]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.76, 95% CI 2-sided [0.79 to 2.72]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.13, 95% CI 2-sided [0.47 to 1.79]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; p = 0.021, ANOVA; LS Mean difference = 0.76, 95% CI 2-sided [0.11 to 1.41]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 8]; Test type: Superiority or Other; p = 0.027, ANOVA; LS Mean difference = 0.75, 95% CI 2-sided [0.09 to 1.41]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 1 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.75, 95% CI 2-sided [3.65 to 5.84]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.21, 95% CI 2-sided [3.13 to 5.29]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.47, 95% CI 2-sided [3.37 to 5.56]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.92, 95% CI 2-sided [2.83 to 5.02]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p = 0.031, ANOVA; LS Mean difference = 0.83, 95% CI 2-sided [0.08 to 1.58]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p = 0.442, ANOVA; LS Mean difference = 0.29, 95% CI 2-sided [-0.44 to 1.02]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 15]; Test type: Superiority or Other; p = 0.152, ANOVA; LS Mean difference = 0.55, 95% CI 2-sided [-0.20 to 1.30]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 1.5 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.62, 95% CI 2-sided [4.52 to 6.72]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.04, 95% CI 2-sided [3.96 to 6.13]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.40, 95% CI 2-sided [4.30 to 6.50]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.88, 95% CI 2-sided [3.78 to 5.98]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.055, ANOVA; LS Mean difference = 0.74, 95% CI 2-sided [-0.01 to 1.49]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.666, ANOVA; LS Mean difference = 0.16, 95% CI 2-sided [-0.57 to 0.90]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 22]; Test type: Superiority or Other; p = 0.181, ANOVA; LS Mean difference = 0.51, 95% CI 2-sided [-0.24 to 1.27]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 2 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.86, 95% CI 2-sided [4.71 to 7.01]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.43, 95% CI 2-sided [4.29 to 6.57]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.79, 95% CI 2-sided [4.64 to 6.94]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.34, 95% CI 2-sided [4.19 to 6.50]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; p = 0.200, ANOVA; LS Mean difference = 0.52, 95% CI 2-sided [-0.27 to 1.31]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; p = 0.831, ANOVA; LS Mean difference = 0.08, 95% CI 2-sided [-0.69 to 0.85]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 29]; Test type: Superiority or Other; p = 0.268, ANOVA; LS Mean difference = 0.45, 95% CI 2-sided [-0.34 to 1.24]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 3 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.73, 95% CI 2-sided [4.54 to 6.91]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.31, 95% CI 2-sided [4.13 to 6.48]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.60, 95% CI 2-sided [4.41 to 6.78]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.35, 95% CI 2-sided [4.17 to 6.54]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; p = 0.367, ANOVA; LS Mean difference = 0.37, 95% CI 2-sided [-0.44 to 1.19]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; p = 0.908, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.84 to 0.75]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 36]; Test type: Superiority or Other; p = 0.553, ANOVA; LS Mean difference = 0.25, 95% CI 2-sided [-0.57 to 1.06]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 4 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.45, 95% CI 2-sided [4.22 to 6.68]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.10, 95% CI 2-sided [3.88 to 6.31]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.42, 95% CI 2-sided [4.19 to 6.66]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.17, 95% CI 2-sided [3.94 to 6.40]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p = 0.518, ANOVA; LS Mean difference = 0.28, 95% CI 2-sided [-0.57 to 1.12]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p = 0.860, ANOVA; LS Mean difference = -0.07, 95% CI 2-sided [-0.90 to 0.75]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 43]; Test type: Superiority or Other; p = 0.556, ANOVA; LS Mean difference = 0.25, 95% CI 2-sided [-0.59 to 1.10]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 5 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.44, 95% CI 2-sided [4.17 to 6.71]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.93, 95% CI 2-sided [3.68 to 6.19]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.27, 95% CI 2-sided [4.00 to 6.54]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 5.06, 95% CI 2-sided [3.79 to 6.34]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 50]; Test type: Superiority or Other; p = 0.392, ANOVA; LS Mean difference = 0.38, 95% CI 2-sided [-0.49 to 1.25]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 50]; Test type: Superiority or Other; p = 0.762, ANOVA; LS Mean difference = -0.13, 95% CI 2-sided [-0.98 to 0.72]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 50]; Test type: Superiority or Other; p = 0.638, ANOVA; LS Mean difference = 0.21, 95% CI 2-sided [-0.66 to 1.08]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 6 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.55, 95% CI 2-sided [3.20 to 5.90]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.45, 95% CI 2-sided [3.11 to 5.78]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.91, 95% CI 2-sided [3.56 to 6.26]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.39, 95% CI 2-sided [3.04 to 5.74]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 57]; Test type: Superiority or Other; p = 0.741, ANOVA; LS Mean difference = 0.16, 95% CI 2-sided [-0.77 to 1.08]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 57]; Test type: Superiority or Other; p = 0.907, ANOVA; LS Mean difference = 0.05, 95% CI 2-sided [-0.85 to 0.95]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 57]; Test type: Superiority or Other; p = 0.274, ANOVA; LS Mean difference = 0.51, 95% CI 2-sided [-0.41 to 1.44]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 7 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.77, 95% CI 2-sided [2.40 to 5.13]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.91, 95% CI 2-sided [2.56 to 5.26]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.12, 95% CI 2-sided [2.75 to 5.48]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.01, 95% CI 2-sided [2.64 to 5.38]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 64]; Test type: Superiority or Other; p = 0.607, ANOVA; LS Mean difference = -0.25, 95% CI 2-sided [-1.18 to 0.69]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 64]; Test type: Superiority or Other; p = 0.824, ANOVA; LS Mean difference = -0.10, 95% CI 2-sided [-1.02 to 0.81]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 64]; Test type: Superiority or Other; p = 0.827, ANOVA; LS Mean difference = 0.10, 95% CI 2-sided [-0.83 to 1.04]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 8 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.98, 95% CI 2-sided [1.58 to 4.39]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.27, 95% CI 2-sided [1.88 to 4.65]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.12, 95% CI 2-sided [1.71 to 4.52]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.57, 95% CI 2-sided [2.16 to 4.98]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 71]; Test type: Superiority or Other; p = 0.232, ANOVA; LS Mean difference = -0.59, 95% CI 2-sided [-1.55 to 0.38]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 71]; Test type: Superiority or Other; p = 0.522, ANOVA; LS Mean difference = -0.31, 95% CI 2-sided [-1.24 to 0.63]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 71]; Test type: Superiority or Other; p = 0.356, ANOVA; LS Mean difference = -0.45, 95% CI 2-sided [-1.41 to 0.51]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 9 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean difference = 2.31, 95% CI 2-sided [0.92 to 3.69]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.45, 95% CI 2-sided [1.08 to 3.82]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.70, 95% CI 2-sided [1.31 to 4.08]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.85, 95% CI 2-sided [1.46 to 4.23]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 78]; Test type: Superiority or Other; p = 0.264, ANOVA; LS Mean difference = -0.54, 95% CI 2-sided [-1.49 to 0.41]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 78]; Test type: Superiority or Other; p = 0.400, ANOVA; LS Mean difference = -0.40, 95% CI 2-sided [-1.32 to 0.53]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 78]; Test type: Superiority or Other; p = 0.758, ANOVA; LS Mean difference = -0.15, 95% CI 2-sided [-1.10 to 0.80]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 10 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.018, ANOVA; LS Mean difference = 1.62, 95% CI 2-sided [0.27 to 2.97]
Statistical Analysis 86: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p = 0.006, ANOVA; LS Mean difference = 1.88, 95% CI 2-sided [0.55 to 3.21]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.29, 95% CI 2-sided [0.94 to 3.63]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.40, 95% CI 2-sided [1.05 to 3.75]
Statistical Analysis 89: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p = 0.097, ANOVA; LS Mean difference = -0.78, 95% CI 2-sided [-1.70 to 0.14]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p = 0.254, ANOVA; LS Mean difference = -0.52, 95% CI 2-sided [-1.42 to 0.38]
Statistical Analysis 91: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 85]; Test type: Superiority or Other; p = 0.812, ANOVA; LS Mean difference = -0.11, 95% CI 2-sided [-1.03 to 0.81]
Statistical Analysis 92: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 11 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.045, ANOVA; LS Mean difference = 1.32, 95% CI 2-sided [0.03 to 2.61]
Statistical Analysis 93: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 92]; Test type: Superiority or Other; p = 0.015, ANOVA; LS Mean difference = 1.59, 95% CI 2-sided [0.31 to 2.87]
Statistical Analysis 94: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 92]; Test type: Superiority or Other; p = 0.009, ANOVA; LS Mean difference = 1.73, 95% CI 2-sided [0.43 to 3.02]
Statistical Analysis 95: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 92]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 2.08, 95% CI 2-sided [0.78 to 3.37]
Statistical Analysis 96: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 92]; Test type: Superiority or Other; p = 0.094, ANOVA; LS Mean difference = -0.76, 95% CI 2-sided [-1.64 to 0.13]
Statistical Analysis 97: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 92]; Test type: Superiority or Other; p = 0.269, ANOVA; LS Mean difference = -0.49, 95% CI 2-sided [-1.35 to 0.38]
Statistical Analysis 98: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 92]; Test type: Superiority or Other; p = 0.437, ANOVA; LS Mean difference = -0.35, 95% CI 2-sided [-1.23 to 0.53]
Statistical Analysis 99: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 12 hour: Treatment difference and 95% CI were based on LSM from ANOVA with treatment, baseline categorical PSR, baseline numerical PSR, gender and treatment-by-baseline categorical PSR terms used as covariates; Test type: Superiority or Other; p = 0.218, ANOVA; LS Mean difference = 0.74, 95% CI 2-sided [-0.44 to 1.92]
Statistical Analysis 100: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 99]; Test type: Superiority or Other; p = 0.046, ANOVA; LS Mean difference = 1.19, 95% CI 2-sided [0.02 to 2.35]
Statistical Analysis 101: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 6, analysis 99]; Test type: Superiority or Other; p = 0.030, ANOVA; LS Mean difference = 1.31, 95% CI 2-sided [0.13 to 2.49]
Statistical Analysis 102: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 99]; Test type: Superiority or Other; p = 0.004, ANOVA; LS Mean difference = 1.75, 95% CI 2-sided [0.57 to 2.93]
Statistical Analysis 103: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 99]; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean difference = -1.01, 95% CI 2-sided [-1.82 to -0.20]
Statistical Analysis 104: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 99]; Test type: Superiority or Other; p = 0.160, ANOVA; LS Mean difference = -0.56, 95% CI 2-sided [-1.35 to 0.22]
Statistical Analysis 105: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 6, analysis 99]; Test type: Superiority or Other; p = 0.284, ANOVA; LS Mean difference = -0.44, 95% CI 2-sided [-1.25 to 0.37]

7. Secondary Outcome: Sum of Pain Relief Rating and Pain Intensity Difference on 4-Point Categorical Scale (PRID4)
Description: PRID4: sum of PID and PRR at each post-dose time points up to 12 hours. Score range for PRID: -1(worst score) to 7(best score). PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [no pain] to 3 [worst possible pain]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID4: -1 (worst score) to 3 (best score). PRR was assessed on a 5-point categorical pain relief rating scale which ranges from 0 =no relief to 4 =complete relief.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0.25 hour | 0.3 (0.6) | 1.0 (1.3) | 0.7 (1.1) | 1.0 (1.4) | 0.6 (1.0)
  0.5 hour | 0.3 (0.9) | 2.6 (1.8) | 2.2 (1.9) | 2.4 (1.8) | 1.6 (1.4)
  1 hour | 0.5 (1.1) | 4.0 (1.8) | 3.6 (1.8) | 3.9 (1.9) | 3.2 (1.9)
  1.5 hour | 0.5 (1.4) | 4.5 (1.7) | 4.1 (2.0) | 4.5 (1.8) | 3.9 (1.9)
  2 hour | 0.4 (1.4) | 4.6 (1.8) | 4.3 (2.1) | 4.7 (1.9) | 4.2 (2.1)
  3 hour | 0.6 (1.8) | 4.6 (1.8) | 4.4 (2.2) | 4.7 (2.0) | 4.3 (2.2)
  4 hour | 0.7 (1.9) | 4.5 (1.8) | 4.3 (2.3) | 4.6 (2.0) | 4.2 (2.3)
  5 hour | 0.6 (1.9) | 4.3 (1.9) | 4.1 (2.4) | 4.4 (2.3) | 4.1 (2.3)
  6 hour | 0.8 (2.0) | 3.8 (2.2) | 3.9 (2.4) | 4.2 (2.4) | 3.7 (2.5)
  7 hour | 0.7 (2.0) | 3.3 (2.3) | 3.4 (2.4) | 3.6 (2.4) | 3.3 (2.5)
  8 hour | 0.7 (2.0) | 2.7 (2.4) | 2.9 (2.3) | 2.8 (2.4) | 3.0 (2.5)
  9 hour | 0.8 (2.0) | 2.2 (2.4) | 2.2 (2.3) | 2.5 (2.3) | 2.5 (2.4)
  10 hour | 0.8 (2.2) | 1.7 (2.3) | 1.7 (2.2) | 2.2 (2.3) | 2.1 (2.4)
  11 hour | 0.9 (2.3) | 1.4 (2.3) | 1.5 (2.2) | 1.9 (2.2) | 1.9 (2.4)
  12 hour | 0.9 (2.4) | 1.1 (2.0) | 1.2 (2.0) | 1.6 (2.1) | 1.7 (2.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.014, ANOVA; LS mean difference = 0.62, 95% CI 2-sided [0.13 to 1.10]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.066, ANOVA; LS Mean difference = 0.46, 95% CI 2-sided [-0.03 to 0.94]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.004, ANOVA; LS Mean difference = 0.71, 95% CI 2-sided [0.22 to 1.20]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.232, ANOVA; LS Mean difference = 0.30, 95% CI 2-sided [-0.19 to 0.78]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.067, ANOVA; LS Mean difference = 0.32, 95% CI 2-sided [-0.02 to 0.66]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.354, ANOVA; LS Mean difference = 0.16, 95% CI 2-sided [-0.18 to 0.50]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.017, ANOVA; LS Mean difference = 0.42, 95% CI 2-sided [0.08 to 0.76]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.15, 95% CI 2-sided [1.45 to 2.86]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.93, 95% CI 2-sided [1.23 to 2.64]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.09, 95% CI 2-sided [1.39 to 2.80]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.32, 95% CI 2-sided [0.61 to 2.02]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 0.83, 95% CI 2-sided [0.34 to 1.33]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean difference = 0.62, 95% CI 2-sided [0.12 to 1.11]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 8]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 0.77, 95% CI 2-sided [0.28 to 1.27]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.45, 95% CI 2-sided [2.69 to 4.22]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.13, 95% CI 2-sided [2.36 to 3.89]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.49, 95% CI 2-sided [2.72 to 4.26]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.78, 95% CI 2-sided [2.02 to 3.54]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean difference = 0.67, 95% CI 2-sided [0.14 to 1.21]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.202, ANOVA; LS Mean difference = 0.35, 95% CI 2-sided [-0.19 to 0.88]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 15]; Test type: Superiority or Other; p = 0.010, ANOVA; LS Mean difference = 0.71, 95% CI 2-sided [0.17 to 1.24]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.00, 95% CI 2-sided [3.24 to 4.76]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.55, 95% CI 2-sided [2.79 to 4.31]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.03, 95% CI 2-sided [3.27 to 4.79]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.48, 95% CI 2-sided [2.72 to 4.24]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.056, ANOVA; LS Mean difference = 0.52, 95% CI 2-sided [-0.01 to 1.05]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.789, ANOVA; LS Mean difference = 0.07, 95% CI 2-sided [-0.46 to 0.60]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 22]; Test type: Superiority or Other; p = 0.042, ANOVA; LS Mean difference = 0.55, 95% CI 2-sided [0.02 to 1.08]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.17, 95% CI 2-sided [3.37 to 4.98]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.86, 95% CI 2-sided [3.06 to 4.66]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.34, 95% CI 2-sided [3.54 to 5.14]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.89, 95% CI 2-sided [3.09 to 4.69]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.317, ANOVA; LS Mean difference = 0.29, 95% CI 2-sided [-0.28 to 0.85]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.922, ANOVA; LS Mean difference = -0.03, 95% CI 2-sided [-0.59 to 0.53]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 29]; Test type: Superiority or Other; p = 0.112, ANOVA; LS Mean difference = 0.45, 95% CI 2-sided [-0.11 to 1.02]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.10, 95% CI 2-sided [3.27 to 4.94]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.76, 95% CI 2-sided [2.92 to 4.59]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.15, 95% CI 2-sided [3.32 to 4.99]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.89, 95% CI 2-sided [3.05 to 4.72]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.464, ANOVA; LS Mean difference = 0.22, 95% CI 2-sided [-0.37 to 0.81]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.667, ANOVA; LS Mean difference = -0.13, 95% CI 2-sided [-0.71 to 0.45]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 36]; Test type: Superiority or Other; p = 0.368, ANOVA; LS Mean difference = 0.27, 95% CI 2-sided [-0.32 to 0.86]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.94, 95% CI 2-sided [3.08 to 4.81]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.63, 95% CI 2-sided [2.77 to 4.49]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 4.06, 95% CI 2-sided [3.19 to 4.92]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.68, 95% CI 2-sided [2.82 to 4.54]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.397, ANOVA; LS Mean difference = 0.26, 95% CI 2-sided [-0.34 to 0.86]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.866, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.65 to 0.55]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 43]; Test type: Superiority or Other; p = 0.226, ANOVA; LS Mean difference = 0.37, 95% CI 2-sided [-0.23 to 0.97]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.80, 95% CI 2-sided [2.90 to 4.70]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.37, 95% CI 2-sided [2.47 to 4.26]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.89, 95% CI 2-sided [2.99 to 4.79]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.60, 95% CI 2-sided [2.70 to 4.50]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.536, ANOVA; LS Mean difference = 0.20, 95% CI 2-sided [-0.43 to 0.83]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.467, ANOVA; LS Mean difference = -0.23, 95% CI 2-sided [-0.86 to 0.39]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 50]; Test type: Superiority or Other; p = 0.361, ANOVA; LS Mean difference = 0.29, 95% CI 2-sided [-0.34 to 0.92]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.17, 95% CI 2-sided [2.21 to 4.13]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.99, 95% CI 2-sided [2.04 to 3.95]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.51, 95% CI 2-sided [2.55 to 4.47]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 3.04, 95% CI 2-sided [2.09 to 4.00]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.704, ANOVA; LS Mean difference = 0.13, 95% CI 2-sided [-0.54 to 0.80]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.890, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.71 to 0.62]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 57]; Test type: Superiority or Other; p = 0.170, ANOVA; LS Mean difference = 0.47, 95% CI 2-sided [-0.20 to 1.14]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.69, 95% CI 2-sided [1.72 to 3.67]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.58, 95% CI 2-sided [1.61 to 3.56]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.99, 95% CI 2-sided [2.01 to 3.97]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.75, 95% CI 2-sided [1.77 to 3.72]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.882, ANOVA; LS Mean difference = -0.05, 95% CI 2-sided [-0.74 to 0.63]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.640, ANOVA; LS Mean difference = -0.16, 95% CI 2-sided [-0.84 to 0.52]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 64]; Test type: Superiority or Other; p = 0.482, ANOVA; LS Mean difference = 0.24, 95% CI 2-sided [-0.44 to 0.93]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.06, 95% CI 2-sided [1.07 to 3.06]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.17, 95% CI 2-sided [1.17 to 3.16]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.24, 95% CI 2-sided [1.25 to 3.24]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 2.42, 95% CI 2-sided [1.43 to 3.41]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.314, ANOVA; LS Mean difference = -0.36, 95% CI 2-sided [-1.05 to 0.34]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.469, ANOVA; LS Mean difference = -0.25, 95% CI 2-sided [-0.95 to 0.44]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 71]; Test type: Superiority or Other; p = 0.616, ANOVA; LS Mean difference = -0.18, 95% CI 2-sided [-0.87 to 0.52]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 1.57, 95% CI 2-sided [0.57 to 2.56]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.002, ANOVA; LS Mean difference = 1.54, 95% CI 2-sided [0.55 to 2.53]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.95, 95% CI 2-sided [0.95 to 2.94]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p < 0.001, ANOVA; LS Mean difference = 1.91, 95% CI 2-sided [0.92 to 2.90]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.330, ANOVA; LS Mean difference = -0.34, 95% CI 2-sided [-1.04 to 0.35]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.288, ANOVA; LS Mean difference = -0.37, 95% CI 2-sided [-1.06 to 0.32]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 78]; Test type: Superiority or Other; p = 0.916, ANOVA; LS Mean difference = 0.04, 95% CI 2-sided [-0.66 to 0.73]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.041, ANOVA; LS Mean difference = 1.01, 95% CI 2-sided [0.04 to 1.98]
Statistical Analysis 86: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.034, ANOVA; LS Mean difference = 1.05, 95% CI 2-sided [0.08 to 2.01]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.001, ANOVA; LS Mean difference = 1.59, 95% CI 2-sided [0.62 to 2.56]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.003, ANOVA; LS Mean difference = 1.48, 95% CI 2-sided [0.52 to 2.45]
Statistical Analysis 89: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.171, ANOVA; LS Mean difference = -0.47, 95% CI 2-sided [-1.15 to 0.20]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.201, ANOVA; LS Mean difference = -0.44, 95% CI 2-sided [-1.11 to 0.23]
Statistical Analysis 91: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 85]; Test type: Superiority or Other; p = 0.763, ANOVA; LS Mean difference = 0.10, 95% CI 2-sided [-0.57 to 0.78]
Statistical Analysis 92: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.175, ANOVA; LS Mean difference = 0.66, 95% CI 2-sided [-0.30 to 1.61]
Statistical Analysis 93: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.120, ANOVA; LS Mean difference = 0.75, 95% CI 2-sided [-0.20 to 1.70]
Statistical Analysis 94: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.014, ANOVA; LS Mean difference = 1.19, 95% CI 2-sided [0.24 to 2.15]
Statistical Analysis 95: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.007, ANOVA; LS Mean difference = 1.31, 95% CI 2-sided [0.36 to 2.26]
Statistical Analysis 96: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.054, ANOVA; LS Mean difference = -0.66, 95% CI 2-sided [-1.32 to 0.01]
Statistical Analysis 97: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.096, ANOVA; LS Mean difference = -0.56, 95% CI 2-sided [-1.22 to 0.10]
Statistical Analysis 98: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 92]; Test type: Superiority or Other; p = 0.724, ANOVA; LS Mean difference = -0.12, 95% CI 2-sided [-0.79 to 0.55]
Statistical Analysis 99: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.345, ANOVA; LS Mean difference = 0.42, 95% CI 2-sided [-0.46 to 1.30]
Statistical Analysis 100: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.228, ANOVA; LS Mean difference = 0.54, 95% CI 2-sided [-0.34 to 1.41]
Statistical Analysis 101: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.045, ANOVA; LS Mean difference = 0.90, 95% CI 2-sided [0.02 to 1.78]
Statistical Analysis 102: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.016, ANOVA; LS Mean difference = 1.08, 95% CI 2-sided [0.21 to 1.96]
Statistical Analysis 103: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.036, ANOVA; LS Mean difference = -0.66, 95% CI 2-sided [-1.27 to -0.04]
Statistical Analysis 104: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.081, ANOVA; LS Mean difference = -0.54, 95% CI 2-sided [-1.15 to 0.07]
Statistical Analysis 105: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 4, analysis 99]; Test type: Superiority or Other; p = 0.556, ANOVA; LS Mean difference = -0.18, 95% CI 2-sided [-0.80 to 0.43]

8. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference on 4-Point Categorical Scale (SPID4) Over 2, 6, 8 and 12 Hours Post-Dose
Description: Pain intensity was assessed on a 4-point categorical pain severity rating scale. SPID4: Time-weighted sum of PID over post-dose time points. SPID4 score range was -2 (worst score) to 6 (best score) for SPID 0-2, -6 (worst score) to 18 (best score) for SPID 0-6, -8 (worst score) to 24 (best score) for SPID 0-8, -12 (worst score) to 36 (best score) for SPID 0-12. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 [none] to 3 [severe]) from the baseline pain intensity scores (score range: 2 =moderate pain to 3 = severe pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -1 (worst score) to 3 (best score).
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 8 hours, 0 to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0 to 2 hours | 0.1 (1.0) | 2.7 (1.5) | 2.4 (1.5) | 2.7 (1.4) | 2.2 (1.4)
  0 to 6 hours | 0.7 (4.4) | 9.1 (4.5) | 8.5 (5.4) | 9.3 (5.0) | 8.2 (4.9)
  0 to 8 hours | 1.0 (6.1) | 11.2 (6.1) | 10.7 (7.2) | 11.6 (6.6) | 10.4 (6.7)
  0 to 12 hours | 2.0 (10.0) | 13.3 (8.8) | 12.9 (9.9) | 14.1 (9.1) | 13.0 (9.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0-2 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline categorical PSR, treatment-by-baseline categorical PSR and gender terms used as covariates. Statistical testing was done at 5% significance level; LS mean difference = 2.53, 95% CI 2-sided [2.01 to 3.05]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-2 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 2.23, 95% CI 2-sided [1.72 to 2.75]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 0-2 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 2.56, 95% CI 2-sided [2.04 to 3.08]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; 0-2 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 2.09, 95% CI 2-sided [1.57 to 2.60]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-2 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.016, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.44, 95% CI 2-sided [0.08 to 0.81]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-2 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.428, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.14, 95% CI 2-sided [-0.21 to 0.50]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-2 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.47, 95% CI 2-sided [0.11 to 0.84]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0-6 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 8.38, 95% CI 2-sided [6.59 to 10.18]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-6 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 7.68, 95% CI 2-sided [5.89 to 9.47]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 0-6 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 8.70, 95% CI 2-sided [6.91 to 10.50]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; 0-6 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 7.65, 95% CI 2-sided [5.86 to 9.44]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-6 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.250, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.74, 95% CI 2-sided [-0.52 to 1.99]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-6 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.956, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.04, 95% CI 2-sided [-1.21 to 1.28]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-6 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.099, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.06, 95% CI 2-sided [-0.20 to 2.31]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0-8 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 10.22, 95% CI 2-sided [7.78 to 12.66]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-8 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 9.49, 95% CI 2-sided [7.06 to 11.92]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 0-8 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 10.72, 95% CI 2-sided [8.28 to 13.15]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; 0-8 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 9.63, 95% CI 2-sided [7.19 to 12.06]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-8 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.492, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.60, 95% CI 2-sided [-1.11 to 2.30]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-8 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.873, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.14, 95% CI 2-sided [-1.83 to 1.56]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-8 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.210, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.09, 95% CI 2-sided [-0.62 to 2.79]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0-12 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 11.65, 95% CI 2-sided [8.10 to 15.20]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0-12 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 10.94, 95% CI 2-sided [7.40 to 14.48]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 0-12 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 12.65, 95% CI 2-sided [9.10 to 16.20]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; 0-12 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 11.72, 95% CI 2-sided [8.18 to 15.26]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-12 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.957, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.07, 95% CI 2-sided [-2.55 to 2.42]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-12 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.534, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.78, 95% CI 2-sided [-3.25 to 1.69]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0-12 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI were calculated based on LSM from the ANOVA model; Test type: Superiority or Other; p = 0.462, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.93, 95% CI 2-sided [-1.55 to 3.41]

9. Secondary Outcome: Time-weighted Sum of Pain Intensity Difference on 11-Point Numerical Scale (SPID11) Over 2, 6, 8 and 12 Hours Post-Dose
Description: Pain intensity was assessed on an 11-point numerical pain severity rating scale. SPID11: Time-weighted sum of PID scores over 12 hours. SPID11 score range was -10 (worst score) to 20 (best score) for SPID 0-2, -30 (worst score) to 60 (best score) for SPID 0-6, -40 (worst score) to 80 (best score) for SPID 0-8, -60 (worst score) to 120 (best score) for SPID 0-12. PID was calculated by subtracting the pain intensity score at given post-dose time points (pain severity score range: 0 =no pain to 10 =worst possible pain) from the baseline pain intensity scores (score range: 5 =moderate pain to 10 =worst possible pain; as participants with baseline pain score of at least moderate were included in study). Total possible score range for PID: -5 (worst score) to 10 (best score).
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 8 hours, 0 to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0 to 2 hours | 0.1 (2.4) | 8.8 (4.3) | 8.0 (4.5) | 8.6 (4.0) | 7.2 (4.3)
  0 to 6 hours | 1.1 (11.8) | 29.9 (13.0) | 28.8 (16.1) | 30.1 (14.4) | 26.8 (15.0)
  0 to 8 hours | 1.8 (16.8) | 36.9 (17.3) | 36.5 (21.5) | 37.6 (19.3) | 34.2 (20.3)
  0 to12 hours | 4.1 (28.7) | 44.0 (25.0) | 44.5 (29.7) | 46.5 (27.3) | 43.7 (29.2)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — p-value was calculated using ANOVA model with treatment, baseline categorical PSR, treatment-by-baseline categorical PSR, baseline numerical PSR and gender terms used as covariates. Statistical testing was done at 5% significance level; LS mean difference = 9.06, 95% CI 2-sided [7.23 to 10.89]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 8.14, 95% CI 2-sided [6.33 to 9.95]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 8.66, 95% CI 2-sided [6.83 to 10.49]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 7.61, 95% CI 2-sided [5.78 to 9.44]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.024, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 1.45, 95% CI 2-sided [0.19 to 2.70]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; p = 0.392, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 0.53, 95% CI 2-sided [-0.69 to 1.76]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.101, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 1.05, 95% CI 2-sided [-0.21 to 2.30]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 30.23, 95% CI 2-sided [23.97 to 36.48]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 27.93, 95% CI 2-sided [21.74 to 34.11]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 29.86, 95% CI 2-sided [23.60 to 36.12]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 27.59, 95% CI 2-sided [21.33 to 33.86]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 12]; Test type: Superiority or Other; p = 0.228, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 2.63, 95% CI 2-sided [-1.65 to 6.92]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.875, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 0.33, 95% CI 2-sided [-3.84 to 4.51]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 14]; Test type: Superiority or Other; p = 0.299, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 2.27, 95% CI 2-sided [-2.02 to 6.55]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 36.98, 95% CI 2-sided [28.48 to 45.47]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 35.10, 95% CI 2-sided [26.70 to 43.50]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 17]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 37.09, 95% CI 2-sided [28.60 to 45.59]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 18]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 35.17, 95% CI 2-sided [26.67 to 43.68]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.543, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 1.80, 95% CI 2-sided [-4.02 to 7.63]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 20]; Test type: Superiority or Other; p = 0.979, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = -0.07, 95% CI 2-sided [-5.75 to 5.60]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 21]; Test type: Superiority or Other; p = 0.517, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 1.92, 95% CI 2-sided [-3.90 to 7.74]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 42.96, 95% CI 2-sided [30.51 to 55.41]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 23]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 42.20, 95% CI 2-sided [29.90 to 54.51]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 24]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 45.12, 95% CI 2-sided [32.67 to 57.57]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 44.25, 95% CI 2-sided [31.79 to 56.71]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 26]; Test type: Superiority or Other; p = 0.767, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = -1.29, 95% CI 2-sided [-9.82 to 7.25]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 27]; Test type: Superiority or Other; p = 0.629, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = -2.04, 95% CI 2-sided [-10.36 to 6.27]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; p = 0.841, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 0.87, 95% CI 2-sided [-7.66 to 9.39]

10. Secondary Outcome: Time-weighted Sum of Pain Relief Rating (TOTPAR) Over 2, 6, 8, 12 Hours Post-Dose
Description: TOTPAR: time-weighted sum of PRR scores over 2, 6, 8 and 12 hours. TOTPAR score range was 0 (worst score) to 8 (best score) for TOTPAR 0-2, 0 (worst score) to 24 (best score) for TOTPAR 0-6, 0 (worst score) to 32 (best score) for TOTPAR 0-8, 0 (worst score) to 48 (best score) for TOTPAR 0-12. PRR was assessed on a 5-point categorical pain relief rating scale where 0= No relief to 4= Complete relief.
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 8 hours, 0 to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0 to 2 hours | 0.7 (1.1) | 4.7 (1.7) | 4.3 (1.9) | 4.7 (1.8) | 4.0 (1.8)
  0 to 6 hours | 2.8 (5.4) | 15.7 (5.2) | 14.8 (6.5) | 16.0 (6.3) | 14.3 (6.7)
  0 to 8 hours | 4.0 (7.6) | 19.6 (7.2) | 18.9 (8.8) | 20.2 (8.6) | 18.4 (9.2)
  0 to 12 hours | 6.4 (12.6) | 23.9 (11.2) | 23.4 (12.6) | 25.8 (12.9) | 23.9 (13.8)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS mean difference = 3.97, 95% CI 2-sided [3.22 to 4.73]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 3.64, 95% CI 2-sided [2.88 to 4.39]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 4.07, 95% CI 2-sided [3.32 to 4.83]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 3.39, 95% CI 2-sided [2.64 to 4.14]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.031, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.58, 95% CI 2-sided [0.05 to 1.11]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; p = 0.360, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.24, 95% CI 2-sided [-0.28 to 0.77]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.011, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.68, 95% CI 2-sided [0.15 to 1.21]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 13.14, 95% CI 2-sided [10.54 to 15.73]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 11.94, 95% CI 2-sided [9.35 to 14.52]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 13.54, 95% CI 2-sided [10.95 to 16.13]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 12.04, 95% CI 2-sided [9.45 to 14.63]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 12]; Test type: Superiority or Other; p = 0.235, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.10, 95% CI 2-sided [-0.72 to 2.91]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.910, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.10, 95% CI 2-sided [-1.91 to 1.70]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 14]; Test type: Superiority or Other; p = 0.105, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.50, 95% CI 2-sided [-0.32 to 3.31]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 15]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 16.05, 95% CI 2-sided [12.49 to 19.61]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 16]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 14.88, 95% CI 2-sided [11.33 to 18.43]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 17]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 16.76, 95% CI 2-sided [13.20 to 20.32]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 18]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 15.23, 95% CI 2-sided [11.68 to 18.78]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 19]; Test type: Superiority or Other; p = 0.514, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.83, 95% CI 2-sided [-1.66 to 3.32]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 20]; Test type: Superiority or Other; p = 0.783, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.35, 95% CI 2-sided [-2.82 to 2.13]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 21]; Test type: Superiority or Other; p = 0.227, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.53, 95% CI 2-sided [-0.96 to 4.02]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 18.28, 95% CI 2-sided [12.95 to 23.61]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 23]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 17.30, 95% CI 2-sided [11.99 to 22.61]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 24]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 20.45, 95% CI 2-sided [15.13 to 25.78]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 18.92, 95% CI 2-sided [13.61 to 24.24]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 26]; Test type: Superiority or Other; p = 0.736, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.64, 95% CI 2-sided [-4.37 to 3.09]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 27]; Test type: Superiority or Other; p = 0.390, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -1.62, 95% CI 2-sided [-5.32 to 2.08]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; p = 0.420, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.53, 95% CI 2-sided [-2.19 to 5.26]

11. Secondary Outcome: Time-weighted Sum of Pain Relief Rating and Pain Intensity Difference on 4-Point Categorical Scale (SPRID4) Over 2, 6 and 12 Hours Post Dose
Description: SPRID4: Time-weighted sum of PRR and PID based on 4 point categorical pain severity rating scale (PRID) with score range: -2(worst score) to 14 (best score) for SPRID 0-2, -6 (worst score) to 42 (best score) for SPRID 0-6 and -12 (worst score) to 84 (best score) for SPRID 0-12. PRID: sum of PID and PRR at post-dose time point with score range: -1 (worst score) to 7 (best score). PID calculated by subtracting pain intensity score at post-dose time points (score range: 0 [none] to 3 [severe]) from baseline pain intensity scores (score range: 2 =moderate pain to 3 = severe pain; as participants with baseline score of at least moderate were included). PID total possible score range: -1 (worst score) to 3(best score). PRR assessed on 5-point categorical scale with range: 0 =no relief to 4 =complete relief.
Time Frame: 0 to 2 hours, 0 to 6 hours, 0 to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale
  0 to 2 hours | 0.9 (2.0) | 7.4 (3.0) | 6.7 (3.2) | 7.4 (3.1) | 6.2 (3.1)
  0 to 6 hours | 3.5 (9.4) | 24.8 (9.2) | 23.3 (11.6) | 25.3 (10.9) | 22.5 (11.2)
  0 to 12 hours | 8.4 (22.0) | 37.2 (19.2) | 36.3 (21.9) | 39.9 (21.1) | 36.9 (22.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS mean difference = 6.50, 95% CI 2-sided [5.25 to 7.76]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 2]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 5.87, 95% CI 2-sided [4.62 to 7.11]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 3]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 6.63, 95% CI 2-sided [5.38 to 7.88]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 4]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 5.48, 95% CI 2-sided [4.23 to 6.73]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 5]; Test type: Superiority or Other; p = 0.022, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.03, 95% CI 2-sided [0.15 to 1.90]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 6]; Test type: Superiority or Other; p = 0.380, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 0.39, 95% CI 2-sided [-0.48 to 1.26]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 7]; Test type: Superiority or Other; p = 0.010, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.15, 95% CI 2-sided [0.28 to 2.03]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 8]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 21.52, 95% CI 2-sided [17.17 to 25.87]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 9]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 9, analysis 1]; LS Mean difference = 19.62, 95% CI 2-sided [15.29 to 23.95]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 10]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 22.24, 95% CI 2-sided [17.89 to 26.59]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 11]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 19.69, 95% CI 2-sided [15.35 to 24.02]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 12]; Test type: Superiority or Other; p = 0.237, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 1.83, 95% CI 2-sided [-1.21 to 4.88]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 13]; Test type: Superiority or Other; p = 0.965, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.07, 95% CI 2-sided [-3.09 to 2.95]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 14]; Test type: Superiority or Other; p = 0.099, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 2.56, 95% CI 2-sided [-0.48 to 5.60]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 22]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 29.93, 95% CI 2-sided [21.14 to 38.73]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 23]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 28.24, 95% CI 2-sided [19.48 to 37.00]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 8, analysis 24]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 33.10, 95% CI 2-sided [24.31 to 41.89]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 25]; Test type: Superiority or Other; p < 0.001, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 30.64, 95% CI 2-sided [21.87 to 39.41]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 26]; Test type: Superiority or Other; p = 0.821, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -0.71, 95% CI 2-sided [-6.86 to 5.44]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 27]; Test type: Superiority or Other; p = 0.440, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = -2.40, 95% CI 2-sided [-8.51 to 3.71]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 8, analysis 28]; Test type: Superiority or Other; p = 0.432, ANOVA — [p-value comment as in outcome 8, analysis 1]; LS Mean difference = 2.46, 95% CI 2-sided [-3.69 to 8.61]

12. Secondary Outcome: Cumulative Percentage of Participants With Meaningful Relief
Description: Percentage of participants with meaningful relief was reported. Participants evaluated time to meaningful relief by stopping a second stopwatch labeled "meaningful relief" at the moment they first began to experience meaningful relief. Stopwatch was active up to 12 hours after dosing or until stopped by participant, or participant became treatment failure prior to depressing the second stopwatch. Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
percentage of participants
  0.25 hours | 0.0 | 1.1 | 1.1 | 3.4 | 1.1
  0.5 hours | 0.0 | 33.3 | 23.7 | 22.5 | 13.0
  1 hour | 3.3 | 65.6 | 54.8 | 67.4 | 54.3
  1.5 hours | 6.7 | 81.1 | 69.9 | 77.5 | 66.3
  2 hours | 10.0 | 85.6 | 77.4 | 84.3 | 73.9
  3 hours | 10.0 | 90.0 | 81.7 | 88.8 | 80.4
  4 hours | 13.3 | 90.0 | 83.9 | 89.9 | 81.5
  5 hours | 13.3 | 91.1 | 84.9 | 89.9 | 82.6
  6 hours | 16.7 | 91.1 | 86.0 | 89.9 | 83.7
  7 hours | 16.7 | 91.1 | 87.1 | 89.9 | 84.8
  8 hours | 16.7 | 91.1 | 88.2 | 89.9 | 85.9
  9 hours | 16.7 | 91.1 | 88.2 | 89.9 | 85.9
  10 hours | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  11 hours | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  12 hours | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.25 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and its associated 95% CI was calculated based on Cochran-Mantel-Haenszel (CMH) adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.571, Cochran-Mantel-Haenszel — p-value was calculated using CMH test which was adjusted for baseline PSR and gender terms. Statistical testing was done at 5% significance level; Difference in proportion = 1.08, 95% CI 2-sided [-1.04 to 3.20]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.25 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.593, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 0.98, 95% CI 2-sided [-0.94 to 2.90]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 0.25 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.282, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.65, 95% CI 2-sided [-0.39 to 7.68]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; 0.25 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.552, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.16, 95% CI 2-sided [-1.11 to 3.42]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0.25 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.994, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -0.01, 95% CI 2-sided [-3.13 to 3.11]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0.25 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.879, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -0.23, 95% CI 2-sided [-3.26 to 2.80]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0.25 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.280, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.33, 95% CI 2-sided [-1.98 to 6.64]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.5 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 33.67, 95% CI 2-sided [24.54 to 42.81]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 0.5 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 23.34, 95% CI 2-sided [14.93 to 31.75]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 0.5 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 22.28, 95% CI 2-sided [13.55 to 31.00]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; 0.5 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.035, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 13.39, 95% CI 2-sided [6.28 to 20.50]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0.5 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 20.14, 95% CI 2-sided [8.67 to 31.62]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0.5 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.088, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 9.56, 95% CI 2-sided [-1.39 to 20.51]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 0.5 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.100, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 9.36, 95% CI 2-sided [-1.73 to 20.45]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 1 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 62.54, 95% CI 2-sided [50.93 to 74.15]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 51.66, 95% CI 2-sided [39.50 to 63.82]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 1 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 64.68, 95% CI 2-sided [52.92 to 76.43]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; 1 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 52.03, 95% CI 2-sided [40.43 to 63.63]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 1 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.138, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 10.66, 95% CI 2-sided [-3.04 to 24.35]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 1 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.935, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -0.59, 95% CI 2-sided [-14.71 to 13.52]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 1 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.063, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 13.30, 95% CI 2-sided [-0.57 to 27.17]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 1.5 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.68, 95% CI 2-sided [62.82 to 86.53]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 1.5 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 63.18, 95% CI 2-sided [50.42 to 75.95]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 1.5 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.39, 95% CI 2-sided [59.21 to 83.57]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; 1.5 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 60.50, 95% CI 2-sided [47.89 to 73.11]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 1.5 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.027, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 14.43, 95% CI 2-sided [1.97 to 26.89]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 1.5 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.729, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.35, 95% CI 2-sided [-10.91 to 15.61]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 1.5 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.087, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 11.33, 95% CI 2-sided [-1.55 to 24.21]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 2 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 75.60, 95% CI 2-sided [62.50 to 88.70]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 2 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 67.45, 95% CI 2-sided [53.65 to 81.24]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 2 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.46, 95% CI 2-sided [61.21 to 87.70]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; 2 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 64.23, 95% CI 2-sided [50.30 to 78.17]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 2 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.052, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 11.59, 95% CI 2-sided [0.12 to 23.06]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 2 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.652, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.84, 95% CI 2-sided [-9.49 to 15.16]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 2 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.090, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 10.28, 95% CI 2-sided [-1.47 to 22.03]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 3 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 79.93, 95% CI 2-sided [67.41 to 92.46]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 3 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.65, 95% CI 2-sided [58.25 to 85.05]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 3 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 78.92, 95% CI 2-sided [66.29 to 91.56]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; 3 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 70.56, 95% CI 2-sided [57.04 to 84.07]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 3 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.069, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 9.61, 95% CI 2-sided [-0.59 to 19.80]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 3 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.911, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 0.65, 95% CI 2-sided [-10.73 to 12.03]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 3 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.127, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.27, 95% CI 2-sided [-2.23 to 18.77]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 4 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 76.55, 95% CI 2-sided [62.37 to 90.72]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 4 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 70.60, 95% CI 2-sided [55.93 to 85.28]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 4 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 76.50, 95% CI 2-sided [62.22 to 90.79]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; 4 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.05, 95% CI 2-sided [53.02 to 83.09]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 4 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.098, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.57, 95% CI 2-sided [-1.47 to 18.61]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 4 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.721, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.01, 95% CI 2-sided [-9.02 to 13.04]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 4 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.115, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.28, 95% CI 2-sided [-1.85 to 18.41]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 5 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 77.66, 95% CI 2-sided [63.63 to 91.69]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 5 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.65, 95% CI 2-sided [57.07 to 86.22]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 5 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 76.50, 95% CI 2-sided [62.22 to 90.79]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; 5 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.10, 95% CI 2-sided [54.14 to 84.06]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 5 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.56, 95% CI 2-sided [-1.15 to 18.27]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 5 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.714, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.01, 95% CI 2-sided [-8.76 to 12.77]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 5 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.164, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 7.21, 95% CI 2-sided [-2.80 to 17.22]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 6 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.38, 95% CI 2-sided [59.56 to 89.20]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 6 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.50, 95% CI 2-sided [54.29 to 84.70]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 6 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 73.24, 95% CI 2-sided [58.18 to 88.30]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; 6 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 67.00, 95% CI 2-sided [51.40 to 82.61]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 6 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.129, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 7.46, 95% CI 2-sided [-2.12 to 17.04]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 6 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.712, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.97, 95% CI 2-sided [-8.50 to 12.43]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 6 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.229, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 6.12, 95% CI 2-sided [-3.76 to 16.00]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 7 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.38, 95% CI 2-sided [59.56 to 89.20]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 7 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 70.54, 95% CI 2-sided [55.45 to 85.64]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 7 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 73.24, 95% CI 2-sided [58.18 to 88.30]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; 7 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.05, 95% CI 2-sided [52.53 to 83.57]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 7 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.186, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 6.38, 95% CI 2-sided [-3.05 to 15.81]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 7 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.703, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.97, 95% CI 2-sided [-8.18 to 12.12]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 7 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.312, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.06, 95% CI 2-sided [-4.68 to 14.79]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 8 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.38, 95% CI 2-sided [59.56 to 89.20]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 8 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.59, 95% CI 2-sided [56.61 to 86.57]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 8 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 73.24, 95% CI 2-sided [58.18 to 88.30]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; 8 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.21, 95% CI 2-sided [53.86 to 84.56]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 8 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 8 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 8 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 9 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.38, 95% CI 2-sided [59.56 to 89.20]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 9 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.59, 95% CI 2-sided [56.61 to 86.57]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 9 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 73.24, 95% CI 2-sided [58.18 to 88.30]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; 9 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.21, 95% CI 2-sided [53.86 to 84.56]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 9 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 9 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 9 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 10 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 86: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 10 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 10 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 400 mg; 10 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 89: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 10 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 10 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 91: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 10 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 92: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 11 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 93: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 11 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 94: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 11 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 95: Comparison: Placebo vs Ibuprofen 400 mg; 11 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 96: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 11 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 97: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 11 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 98: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 11 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 99: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 12 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 100: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; 12 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 101: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; 12 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 102: Comparison: Placebo vs Ibuprofen 400 mg; 12 hours: Treatment difference (Ibuprofen 400 mg - placebo) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 103: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 12 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 104: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 12 hours: Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 105: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; 12 hours: Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg) and corresponding 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]

13. Secondary Outcome: Cumulative Percentage of Participants With Confirmed First Perceptible Relief
Description: Percentage of participants with confirmed first perceptible relief was reported. Participants evaluated the time to first perceptible relief (confirmed by meaningful relief) by stopping the first stopwatch labelled 'first perceptible relief' at the moment they first began to experience any pain relief, if the participant also achieved meaningful relief by the end of the study. Stopwatch was active up to 12 hours after dosing or until stopped by the participant, or until the participant dropped out due to treatment failure prior to depressing the first stopwatch or until the time of withdrawal (discontinuation). Treatment failure was defined as participant taking rescue medication, or discontinuing due to lack of efficacy.
Time Frame: 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
percentage of participants
  0.25 hour | 3.3 | 26.7 | 18.3 | 28.1 | 19.6
  0.5 hour | 10.0 | 73.3 | 66.7 | 77.5 | 63.0
  1 hour | 16.7 | 88.9 | 83.9 | 88.8 | 80.4
  1.5 hour | 16.7 | 91.1 | 86.0 | 89.9 | 84.8
  2 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  3 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  4 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  5 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  6 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  7 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  8 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  9 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  10 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  11 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
  12 hour | 20.0 | 91.1 | 88.2 | 89.9 | 85.9
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; 0.25 hours: Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo) and its associated 95% CI was calculated based on CMH adjusted proportions and the corresponding standard error; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 23.99, 95% CI 2-sided [13.32 to 34.67]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 2]; Test type: Superiority or Other; p = 0.048, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 14.83, 95% CI 2-sided [4.59 to 25.07]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 3]; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 24.98, 95% CI 2-sided [13.43 to 36.53]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 4]; Test type: Superiority or Other; p = 0.030, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 16.57, 95% CI 2-sided [6.25 to 26.88]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 5]; Test type: Superiority or Other; p = 0.269, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 6.86, 95% CI 2-sided [-4.80 to 18.53]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 6]; Test type: Superiority or Other; p = 0.735, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -1.95, 95% CI 2-sided [-13.34 to 9.43]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 7]; Test type: Superiority or Other; p = 0.176, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.58, 95% CI 2-sided [-3.88 to 21.04]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 8]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 63.30, 95% CI 2-sided [49.07 to 77.52]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 9]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 56.81, 95% CI 2-sided [42.28 to 71.34]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 10]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 67.57, 95% CI 2-sided [53.58 to 81.55]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 11]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 53.31, 95% CI 2-sided [38.62 to 67.99]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 12]; Test type: Superiority or Other; p = 0.140, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 10.28, 95% CI 2-sided [-3.26 to 23.82]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 13]; Test type: Superiority or Other; p = 0.674, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.98, 95% CI 2-sided [-10.94 to 16.89]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 14]; Test type: Superiority or Other; p = 0.034, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 14.58, 95% CI 2-sided [1.22 to 27.93]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 15]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 72.32, 95% CI 2-sided [58.25 to 86.39]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 16]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 67.20, 95% CI 2-sided [52.63 to 81.78]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 17]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 72.40, 95% CI 2-sided [58.40 to 86.40]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 18]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 64.12, 95% CI 2-sided [49.32 to 78.91]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 19]; Test type: Superiority or Other; p = 0.119, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.40, 95% CI 2-sided [-2.06 to 18.85]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 20]; Test type: Superiority or Other; p = 0.616, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 2.84, 95% CI 2-sided [-8.30 to 13.98]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 21]; Test type: Superiority or Other; p = 0.125, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 8.34, 95% CI 2-sided [-2.20 to 18.87]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 22]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 74.49, 95% CI 2-sided [60.73 to 88.25]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 23]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.38, 95% CI 2-sided [55.05 to 83.71]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 24]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 73.52, 95% CI 2-sided [59.65 to 87.38]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.36, 95% CI 2-sided [54.01 to 82.71]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 26]; Test type: Superiority or Other; p = 0.187, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 6.33, 95% CI 2-sided [-2.99 to 15.65]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 27]; Test type: Superiority or Other; p = 0.881, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 0.79, 95% CI 2-sided [-9.42 to 10.99]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 28]; Test type: Superiority or Other; p = 0.311, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.05, 95% CI 2-sided [-4.60 to 14.71]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 29]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 30]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 32]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 33]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 34]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 35]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 36]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 38]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 39]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 40]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 41]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 42]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 44]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 45]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 46]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 47]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 48]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 49]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 50]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 51]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 52]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 53]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 54]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 55]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 56]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 57]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 58]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 59]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 60]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 61]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 62]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 63]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 64]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 65]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 66]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 68]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 69]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 70]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 71]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 72]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 73]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 74]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 75]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 76]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 77]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 78]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 79]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 80]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 81]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 82]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 83]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 84]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 85: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 85]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 86: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 86]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 87: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 87]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 88: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 88]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 89: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 89]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 90: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 90]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 91: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 91]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 92: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 92]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 93: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 93]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 94: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 94]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 95: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 95]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 96: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 96]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 97: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 97]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 98: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 98]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]
Statistical Analysis 99: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 99]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 71.10, 95% CI 2-sided [55.82 to 86.38]
Statistical Analysis 100: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 100]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 68.31, 95% CI 2-sided [52.88 to 83.74]
Statistical Analysis 101: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 101]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 69.98, 95% CI 2-sided [54.47 to 85.48]
Statistical Analysis 102: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 102]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 65.95, 95% CI 2-sided [50.16 to 81.74]
Statistical Analysis 103: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 103]; Test type: Superiority or Other; p = 0.265, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.25, 95% CI 2-sided [-3.92 to 14.41]
Statistical Analysis 104: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 104]; Test type: Superiority or Other; p = 0.710, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.85, 95% CI 2-sided [-7.82 to 11.53]
Statistical Analysis 105: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 105]; Test type: Superiority or Other; p = 0.416, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 3.99, 95% CI 2-sided [-5.52 to 13.49]

14. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the time interval from the study drug administration up to the first documentation of treatment failure. Treatment failure was defined as taking the rescue medication or discontinuation of the participants from the study due to lack of efficacy, whichever came first. Participants were censored at 12 hours or at their final assessment time, whichever came first.
Time Frame: From 0 hour up to 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
hours | 1.6 [1.3 to 1.8] | 9.7 [8.7 to NA] — Upper limit of confidence interval was not estimable as it was >720 minutes/12 hours) for Ibuprofen 200 mg + Acetaminophen 500 mg group. | 10.1 [9.2 to 12] | 11.1 [9.2 to NA] — Upper limit of confidence interval was not estimable as it was >720 minutes/12 hours) for Ibuprofen 300 mg + Acetaminophen 500 mg group. | 10.4 [9.2 to NA] — Upper limit of confidence interval was not estimable as it was >720 minutes/12 hours) for Ibuprofen 400 mg group.
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - placebo), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p < 0.001, Proportional hazards model — p-value was calculated using PH model with treatment, baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.17 to 0.45]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - placebo), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 14, analysis 1]; LS mean difference = 0.24, 95% CI 2-sided [0.15 to 0.39]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - placebo), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 14, analysis 1]; LS mean difference = 0.21, 95% CI 2-sided [0.13 to 0.35]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; Treatment difference (Ibuprofen 400 mg - placebo), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p < 0.001, Proportional hazards model — [p-value comment as in outcome 14, analysis 1]; LS mean difference = 0.25, 95% CI 2-sided [0.15 to 0.41]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; Treatment difference (Ibuprofen 200 mg + Acetaminophen 500 mg - Ibuprofen 400 mg), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p = 0.549, Proportional hazards model — [p-value comment as in outcome 14, analysis 1]; LS mean difference = 1.12, 95% CI 2-sided [0.77 to 1.63]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; Treatment difference (Ibuprofen 250 mg + Acetaminophen 500 mg - Ibuprofen 400 mg), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p = 0.863, Proportional hazards model — [p-value comment as in outcome 14, analysis 1]; LS mean difference = 0.97, 95% CI 2-sided [0.66 to 1.42]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; Treatment difference (Ibuprofen 300 mg + Acetaminophen 500 mg - Ibuprofen 400 mg), p-value, HR and corresponding 95% CI were calculated based on the Wald statistic from the PH model with treatment, baseline categorical pain severity rating and gender terms used as covariates; Test type: Superiority or Other; p = 0.454, Proportional hazards model — [p-value comment as in outcome 14, analysis 1]; LS mean difference = 0.86, 95% CI 2-sided [0.57 to 1.28]

15. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: Treatment failure was defined as taking the rescue medication or discontinuation of the participants from the study due to lack of efficacy, whichever came first. Participants were censored at 12 hours or at their final assessment time, whichever came first. Percentage of participants who had treatment failure were reported.
Time Frame: 1.5, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
percentage of participants
  1.5 hour | 43.3 | 2.2 | 2.2 | 4.5 | 5.4
  2 hour | 73.3 | 2.2 | 6.5 | 5.6 | 10.9
  3 hour | 80.0 | 2.2 | 8.6 | 6.7 | 13.0
  4 hour | 80.0 | 3.3 | 9.7 | 7.9 | 15.2
  5 hour | 80.0 | 4.4 | 14.0 | 10.1 | 15.2
  6 hour | 80.0 | 8.9 | 18.3 | 14.6 | 20.7
  7 hour | 80.0 | 17.8 | 20.4 | 15.7 | 27.2
  8 hour | 80.0 | 28.9 | 23.7 | 25.8 | 32.6
  9 hour | 80.0 | 40.0 | 33.3 | 36.0 | 35.9
  10 hour | 80.0 | 51.1 | 46.2 | 42.7 | 45.7
  11 hour | 80.0 | 57.8 | 53.8 | 48.3 | 53.3
  12 hour | 80.0 | 64.4 | 57.0 | 50.6 | 55.4
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 22]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -41.07, 95% CI 2-sided [-59.56 to -22.58]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 23]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -40.98, 95% CI 2-sided [-59.41 to -22.56]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 24]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -38.64, 95% CI 2-sided [-57.49 to -19.79]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 25]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -38.11, 95% CI 2-sided [-56.94 to -19.28]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 26]; Test type: Superiority or Other; p = 0.274, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -3.13, 95% CI 2-sided [-8.67 to 2.40]
Statistical Analysis 6: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 27]; Test type: Superiority or Other; p = 0.304, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -2.89, 95% CI 2-sided [-8.40 to 2.62]
Statistical Analysis 7: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 28]; Test type: Superiority or Other; p = 0.769, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -0.96, 95% CI 2-sided [-7.41 to 5.49]
Statistical Analysis 8: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 29]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -71.19, 95% CI 2-sided [-88.00 to -54.38]
Statistical Analysis 9: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 30]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -66.99, 95% CI 2-sided [-84.26 to -49.72]
Statistical Analysis 10: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 31]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -67.47, 95% CI 2-sided [-84.75 to -50.19]
Statistical Analysis 11: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 32]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -62.76, 95% CI 2-sided [-80.45 to -45.07]
Statistical Analysis 12: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 33]; Test type: Superiority or Other; p = 0.021, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -8.53, 95% CI 2-sided [-15.55 to -1.50]
Statistical Analysis 13: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 34]; Test type: Superiority or Other; p = 0.337, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -3.99, 95% CI 2-sided [-12.05 to 4.07]
Statistical Analysis 14: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 35]; Test type: Superiority or Other; p = 0.204, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -5.26, 95% CI 2-sided [-13.28 to 2.76]
Statistical Analysis 15: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 36]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -77.89, 95% CI 2-sided [-92.29 to -63.49]
Statistical Analysis 16: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 37]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -71.65, 95% CI 2-sided [-86.71 to -56.58]
Statistical Analysis 17: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 38]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -72.87, 95% CI 2-sided [-88.06 to -57.68]
Statistical Analysis 18: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 39]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -67.20, 95% CI 2-sided [-82.87 to -51.52]
Statistical Analysis 19: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 40]; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -10.71, 95% CI 2-sided [-18.20 to -3.21]
Statistical Analysis 20: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 41]; Test type: Superiority or Other; p = 0.385, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -3.99, 95% CI 2-sided [-12.86 to 4.88]
Statistical Analysis 21: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 42]; Test type: Superiority or Other; p = 0.162, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -6.29, 95% CI 2-sided [-14.97 to 2.40]
Statistical Analysis 22: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 43]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -76.81, 95% CI 2-sided [-91.35 to -62.27]
Statistical Analysis 23: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 44]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -70.60, 95% CI 2-sided [-85.79 to -55.41]
Statistical Analysis 24: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 45]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -71.66, 95% CI 2-sided [-87.00 to -56.31]
Statistical Analysis 25: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 46]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -65.19, 95% CI 2-sided [-81.03 to -49.34]
Statistical Analysis 26: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 47]; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -11.70, 95% CI 2-sided [-19.86 to -3.55]
Statistical Analysis 27: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 48]; Test type: Superiority or Other; p = 0.310, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -4.94, 95% CI 2-sided [-14.34 to 4.46]
Statistical Analysis 28: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 49]; Test type: Superiority or Other; p = 0.126, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -7.36, 95% CI 2-sided [-16.63 to 1.90]
Statistical Analysis 29: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 50]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -75.64, 95% CI 2-sided [-90.35 to -60.93]
Statistical Analysis 30: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 51]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -66.43, 95% CI 2-sided [-81.99 to -50.88]
Statistical Analysis 31: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 52]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -69.33, 95% CI 2-sided [-84.96 to -53.71]
Statistical Analysis 32: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 53]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -65.19, 95% CI 2-sided [-81.03 to -49.34]
Statistical Analysis 33: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 54]; Test type: Superiority or Other; p = 0.016, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -10.61, 95% CI 2-sided [-19.02 to -2.19]
Statistical Analysis 34: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 55]; Test type: Superiority or Other; p = 0.895, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -0.69, 95% CI 2-sided [-10.69 to 9.32]
Statistical Analysis 35: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 56]; Test type: Superiority or Other; p = 0.308, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -5.09, 95% CI 2-sided [-14.80 to 4.62]
Statistical Analysis 36: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 57]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -71.36, 95% CI 2-sided [-86.58 to -56.13]
Statistical Analysis 37: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 58]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -62.11, 95% CI 2-sided [-78.04 to -46.19]
Statistical Analysis 38: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 59]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -64.57, 95% CI 2-sided [-80.64 to -48.50]
Statistical Analysis 39: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 60]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -59.84, 95% CI 2-sided [-76.12 to -43.55]
Statistical Analysis 40: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 61]; Test type: Superiority or Other; p = 0.028, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -11.49, 95% CI 2-sided [-21.63 to -1.35]
Statistical Analysis 41: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 62]; Test type: Superiority or Other; p = 0.747, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -1.88, 95% CI 2-sided [-13.15 to 9.38]
Statistical Analysis 42: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 63]; Test type: Superiority or Other; p = 0.303, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -5.88, 95% CI 2-sided [-16.88 to 5.12]
Statistical Analysis 43: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 64]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -62.49, 95% CI 2-sided [-78.64 to -46.34]
Statistical Analysis 44: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 65]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -60.09, 95% CI 2-sided [-76.15 to -44.02]
Statistical Analysis 45: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 66]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -63.45, 95% CI 2-sided [-79.64 to -47.27]
Statistical Analysis 46: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 67]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -53.41, 95% CI 2-sided [-70.10 to -36.72]
Statistical Analysis 47: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 68]; Test type: Superiority or Other; p = 0.137, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -9.14, 95% CI 2-sided [-21.18 to 2.90]
Statistical Analysis 48: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 69]; Test type: Superiority or Other; p = 0.311, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -6.34, 95% CI 2-sided [-18.39 to 5.71]
Statistical Analysis 49: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 70]; Test type: Superiority or Other; p = 0.067, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -11.23, 95% CI 2-sided [-22.97 to 0.52]
Statistical Analysis 50: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 71]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -51.54, 95% CI 2-sided [-68.42 to -34.66]
Statistical Analysis 51: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 72]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -57.01, 95% CI 2-sided [-73.27 to -40.76]
Statistical Analysis 52: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 73]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -53.21, 95% CI 2-sided [-70.16 to -36.26]
Statistical Analysis 53: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 74]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -47.82, 95% CI 2-sided [-64.81 to -30.83]
Statistical Analysis 54: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 75]; Test type: Superiority or Other; p = 0.604, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -3.52, 95% CI 2-sided [-16.89 to 9.85]
Statistical Analysis 55: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 76]; Test type: Superiority or Other; p = 0.184, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -8.78, 95% CI 2-sided [-21.50 to 3.94]
Statistical Analysis 56: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 77]; Test type: Superiority or Other; p = 0.340, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -6.43, 95% CI 2-sided [-19.56 to 6.70]
Statistical Analysis 57: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 78]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -40.27, 95% CI 2-sided [-57.67 to -22.88]
Statistical Analysis 58: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 79]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -47.24, 95% CI 2-sided [-64.21 to -30.27]
Statistical Analysis 59: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 80]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -43.15, 95% CI 2-sided [-60.57 to -25.72]
Statistical Analysis 60: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 81]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -44.45, 95% CI 2-sided [-61.55 to -27.34]
Statistical Analysis 61: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 82]; Test type: Superiority or Other; p = 0.548, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 4.29, 95% CI 2-sided [-9.80 to 18.38]
Statistical Analysis 62: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 83]; Test type: Superiority or Other; p = 0.721, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -2.51, 95% CI 2-sided [-16.20 to 11.18]
Statistical Analysis 63: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 84]; Test type: Superiority or Other; p = 0.951, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 0.44, 95% CI 2-sided [-13.47 to 14.35]
Statistical Analysis 64: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 85]; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -29.13, 95% CI 2-sided [-46.66 to -11.59]
Statistical Analysis 65: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 86]; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -34.30, 95% CI 2-sided [-51.62 to -16.97]
Statistical Analysis 66: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 87]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -36.26, 95% CI 2-sided [-53.80 to -18.73]
Statistical Analysis 67: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 88]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -34.56, 95% CI 2-sided [-51.77 to -17.35]
Statistical Analysis 68: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 89]; Test type: Superiority or Other; p = 0.455, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 5.45, 95% CI 2-sided [-8.89 to 19.79]
Statistical Analysis 69: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 90]; Test type: Superiority or Other; p = 0.953, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 0.43, 95% CI 2-sided [-13.80 to 14.65]
Statistical Analysis 70: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 91]; Test type: Superiority or Other; p = 0.731, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -2.48, 95% CI 2-sided [-16.63 to 11.66]
Statistical Analysis 71: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 92]; Test type: Superiority or Other; p = 0.024, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -22.63, 95% CI 2-sided [-39.97 to -5.29]
Statistical Analysis 72: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 93]; Test type: Superiority or Other; p = 0.009, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -26.87, 95% CI 2-sided [-44.12 to -9.62]
Statistical Analysis 73: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 94]; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -30.76, 95% CI 2-sided [-48.36 to -13.16]
Statistical Analysis 74: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 95]; Test type: Superiority or Other; p = 0.007, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -27.26, 95% CI 2-sided [-44.51 to -10.00]
Statistical Analysis 75: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 96]; Test type: Superiority or Other; p = 0.516, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 4.66, 95% CI 2-sided [-9.50 to 18.82]
Statistical Analysis 76: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 97]; Test type: Superiority or Other; p = 0.939, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 0.55, 95% CI 2-sided [-13.63 to 14.72]
Statistical Analysis 77: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 98]; Test type: Superiority or Other; p = 0.536, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -4.53, 95% CI 2-sided [-18.86 to 9.80]
Statistical Analysis 78: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 99]; Test type: Superiority or Other; p = 0.107, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -15.81, 95% CI 2-sided [-33.02 to 1.41]
Statistical Analysis 79: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 100]; Test type: Superiority or Other; p = 0.019, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -23.71, 95% CI 2-sided [-40.91 to -6.51]
Statistical Analysis 80: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; [analysis description as in outcome 12, analysis 101]; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -28.44, 95% CI 2-sided [-45.99 to -10.88]
Statistical Analysis 81: Comparison: Placebo vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 102]; Test type: Superiority or Other; p = 0.012, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -25.04, 95% CI 2-sided [-42.23 to -7.85]
Statistical Analysis 82: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 103]; Test type: Superiority or Other; p = 0.195, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 9.16, 95% CI 2-sided [-4.75 to 23.08]
Statistical Analysis 83: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 104]; Test type: Superiority or Other; p = 0.835, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = 1.48, 95% CI 2-sided [-12.54 to 15.50]
Statistical Analysis 84: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; [analysis description as in outcome 12, analysis 105]; Test type: Superiority or Other; p = 0.542, Cochran-Mantel-Haenszel — [p-value comment as in outcome 12, analysis 1]; Difference in proportion = -4.41, 95% CI 2-sided [-18.61 to 9.79]

16. Secondary Outcome: Participant Global Evaluation of Study Medication
Description: Participant global evaluation of study medication was performed at the 12-hour time point or immediately before taking the rescue medication. It was scored on a 6-point categorical scale where 0= Very poor, 1= Poor, 2= Fair, 3= Good, 4= Very Good and 5= Excellent.
Time Frame: 12 hour
Population: ITT population included all randomized participants who received study medication and provided a baseline assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Number analyzed (Participants) | 30 | 90 | 93 | 89 | 92
units on a scale | 1.0 (1.5) | 3.8 (1.1) | 3.4 (1.2) | 3.6 (1.2) | 3.5 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen 200 mg + Acetaminophen 500 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — p-value was calculated using CMH test with modified ridit scores, controlling for baseline PSR and gender terms. Statistical testing was done at 5% significance level (2-sided); Mean Difference (Final Values) = 0.90, 95% CI 2-sided [0.79 to 1.01]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen 250 mg + Acetaminophen 500 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = 0.83, 95% CI 2-sided [0.79 to 1.01]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen 300 mg + Acetaminophen 500 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = 0.86, 95% CI 2-sided [0.73 to 0.99]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen 400 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = 0.80, 95% CI 2-sided [0.65 to 0.95]
Statistical Analysis 5: Comparison: Ibuprofen 200 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.174, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.07 to 0.37]
Statistical Analysis 6: Comparison: Ibuprofen 300 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.722, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = 0.04, 95% CI 2-sided [-0.18 to 0.26]
Statistical Analysis 7: Comparison: Ibuprofen 250 mg + Acetaminophen 500 mg vs Ibuprofen 400 mg; Treatment difference and its associated 95% CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.365, Cochran-Mantel-Haenszel — [p-value comment as in outcome 16, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.32 to 0.11]

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen 200 mg + Acetaminophen 500 mg | Ibuprofen 250 mg + Acetaminophen 500 mg | Ibuprofen 300 mg + Acetaminophen 500 mg | Ibuprofen 400 mg
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/90 | 0/93 | 0/89 | 0/92
Other Adverse Events (participants affected / at risk) | 15/30 | 33/90 | 27/93 | 22/89 | 30/92
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=30) | Ibuprofen 200 mg + Acetaminophen 500 mg (N=90) | Ibuprofen 250 mg + Acetaminophen 500 mg (N=93) | Ibuprofen 300 mg + Acetaminophen 500 mg (N=89) | Ibuprofen 400 mg (N=92)
Dizziness (Cardiac disorders) | 3 | 9 | 6 | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Alveolar osteitis (Gastrointestinal disorders) | 0 | 4 | 2 | 1 | 2
Nausea (Gastrointestinal disorders) | 14 | 22 | 18 | 16 | 22
Vomiting (Gastrointestinal disorders) | 7 | 8 | 11 | 5 | 14
Feeling hot (General disorders) | 2 | 4 | 1 | 4 | 4
Hyperhidrosis (General disorders) | 0 | 2 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 4 | 1 | 1 | 4
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 2
Tremor (Nervous system disorders) | 1 | 1 | 2 | 3 | 2
Post procedural haemorrhage (Vascular disorders) | 0 | 0 | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.